CLINICAL TRIAL: NCT03814187
Title: An Open-label Extension Trial of the Phase III Lipid-lowering Trials to Assess the Effect of Long Term Dosing of Inclisiran Given as Subcutaneous Injections in Subjects With High Cardiovascular Risk and Elevated LDL-C
Brief Title: Trial to Assess the Effect of Long Term Dosing of Inclisiran in Subjects With High CV Risk and Elevated LDL-C
Acronym: ORION-8
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDCO-PCS-17-05; CKJX839A12306B (Other: Novartis Pharmaceuticals); 2017-003092-55 (EudraCT Number)
Record Dates: First submitted 2019-01-17; First posted 2019-01-23 (Actual); Results first posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: ASCVD; Elevated Cholesterol; Heterozygous Familial Hypercholesterolemia; Homozygous Familial Hypercholesterolemia
Keywords: Inclisiran sodium; ASCVD; LDL-C; HeFH; HoFH
MeSH Terms: conditions — Hypercholesterolemia; Homozygous Familial Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Inclisiran (Experimental): Inclisiran sodium 300 milligrams (mg) was administered as a single SC injection on Day 1*, 90, then every 180 days to Day 990.
  *Subjects who received blinded placebo in the feeder study received blinded inclisiran and subjects who received blinded inclisiran in the feeder study received blinded placebo on Day 1 in ORION-8. Subjects from the open label ORION-3 study did not receive any injection of study drug on Day 1. Their first dose of study medication was at day 90
  Interventions: Drug: Inclisiran Sodium

INTERVENTIONS:
Drug: Inclisiran Sodium — Inclisiran is a small interfering ribonucleic acid (RNA) that inhibits PCSK9 synthesis.

SUMMARY:
The purpose of this extension study was to evaluate the efficacy, safety, and tolerability of long-term dosing of Inclisiran. The study was a global multicenter study.

DETAILED DESCRIPTION:
This study was an open label, long term extension study in subjects with atherosclerotic cardiovascular disease (ASCVD), ASCVD-risk equivalents (eg, diabetes and familial hypercholesterolemia), or heterozygous familial hypercholesterolemia (HeFH) and elevated low density lipoprotein cholesterol (LDL-C) despite maximum tolerated dose of LDL-C lowering therapies who have completed the inclisiran Phase II trial MDCO-PCS-16-01 (ORION-3; NCT03060577), or any of the following Phase III lipid lowering studies: MDCO-PCS-17-03 (ORION-9; NCT03397121), MDCO-PCS-17-04 (ORION-10; NCT03399370), or MDCO-PCS-17-08 (ORION-11; NCT03400800).

The End of Study (EOS) visit in the previous feeder studies was Day 1 in this extension study.The duration that each subject participated in this study was a maximum of 3 years. However, for subjects from the Study ORION-3, the Sponsor decided to end the study prior to completion of their full 3-year of participation. It is recorded in the database as discontinuation was due to Sponsor's decision.

In this Phase III extension study, the same study drug of inclisiran sodium 300 mg (equivalent to 284 mg inclisiran) was administered as a single subcutaneous (SC) dose every 180 days from the last dose in previous feeder study (except for subjects newly initiating inclisiran, who received the first two doses 90 days apart) until the end of the study.

On Day 1 (EOS visit in the feeder study), subjects from the previous feeder studies received blinded study medication except subjects from Study ORION-3. Subjects who received placebo in the previous Phase III feeder study received blinded inclisiran and subjects who received inclisiran in the previous feeder study received blinded placebo at this visit, so that subjects previously on placebo received the correct dosing regime, i.e. a dose at Day 1, Day 90 and every 180-days thereafter. Subjects previously treated with inclisiran did not need a dose of inclisiran to maintain every 180-dosing regime and therefore, were given placebo in order to maintain the blinding of the feeder study. Subjects that moved over from ORION-3 received the first study medication at Day 90, as this study was already open-label.

On Day 90, all subjects received inclisiran sodium 300 mg. This is 180 days after the last injection in the previous feeder study for subjects that received inclisiran and was the second dose of inclisiran for the subjects that received placebo in the feeder study. The EOS visit occurred at Day 1080.

This extension study allowed subjects continued access to inclisiran treatment and allowed the collection of additional efficacy and safety data for long-term use beyond the end of the feeder studies.

ELIGIBILITY:
Inclusion Criteria:

1. Completion on a previously qualifying inclisiran Phase II trial MDCO-PCS-16-01 (ORION-3), or Phase III lipid lowering ORION feeder study [MDCO-PCS-17-03 (ORION-9), MDCO-PCS-17-4 (ORION-10), or MDCO-PCS-17-08 (ORION-11)] meaning the subject received the last dose of study drug and completed the final study visit per applicable protocol.
2. On current lipid-lowering therapies (such as a statin and/or ezetimibe) from previous study with no planned medication or dose change during study participation.
3. Willing and able to give informed consent before initiation of any study-related procedures and willing to comply with all required study procedures.

Exclusion Criteria:

1. Any uncontrolled or serious disease, or any medical or surgical condition, that may either interfere with participation in the clinical study, and/or put the subject at significant risk [according to investigator's (or delegate's) judgment] if he/she participates in the clinical study.
2. An underlying known disease, or surgical, physical, or medical condition that, in the opinion of the investigator (or delegate) might interfere with interpretation of the clinical study results.
3. Severe concomitant noncardiovascular disease that carries the risk of reducing life expectancy to less than 3 years,
4. Active liver disease defined as any known current infectious, neoplastic, or metabolic pathology of the liver or unexplained alanine aminotransferase (ALT), aspartate aminotransferase (AST), elevation >3x the upper limit of normal (ULN), or total bilirubin (TBIL) elevation >2x ULN at the last recorded visit in the feeder study prior to study entry visit.
5. Females who are pregnant or nursing, or who are of childbearing potential and unwilling to use at least one method of acceptable effective contraception (eg, oral contraceptives, barrier methods, approved contraceptive implant, long-term injectable contraception, intrauterine device) for the entire duration of the study. Exemptions from this criterion:

   1. Women >2 years postmenopausal (defined as 1 year or longer since last menstrual period) and more than 55 years of age.
   2. Postmenopausal women (as defined above) and less than 55 years of age with a negative pregnancy test within 24 hours of randomization.
   3. Women who are surgically sterilized at least 3 months prior to enrollment.
6. Planned use of other investigational medicinal products other than inclisiran or devices during the course of the study.
7. Any condition that according to the investigator could interfere with the conduct of the study, such as but not limited to:

   1. Subjects who are unable to communicate or to cooperate with the investigator
   2. Unable to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study (including subjects whose cooperation is doubtful due to drug abuse or alcohol dependency)
   3. Unlikely to comply with the protocol requirements, instructions, and study-related restrictions (eg, uncooperative attitude, inability to return for follow-up visits, and improbability of completing the study)
   4. Have any medical or surgical condition, which in the opinion of the investigator would put the subject at increased risk from participating in the study
   5. Persons directly involved in the conduct of the study.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3275 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Wright, MD, Principal Investigator — Mayo Clinic
Locations (238):
- United States (141):
  - Research Site 10001-015, Birmingham, Alabama
  - Research Site 10001-138, Foley, Alabama
  - Research Site 10001-113, Huntsville, Alabama
  - Research Site 10001-058, Mobile, Alabama
  - Research Site 10001-037, Montgomery, Alabama
  - Research Site 10001-076, Saraland, Alabama
  - Research Site 10001-013, Chandler, Arizona
  - Research Site 10001-077, Mesa, Arizona
  - Research Site 10001-136, Phoenix, Arizona
  - Research Site 10001-051, Surprise, Arizona
  - Research Site 10001-019, Tucson, Arizona
  - Research Site 10001-004, Tucson, Arizona
  - Research Site 10001-132, Tucson, Arizona
  - Research Site 10001-073, Beverly Hills, California
  - Research Site 10001-050, Canoga Park, California
  - Research Site 10001-011, Carlsbad, California
  - Research Site 10001-065, El Cajon, California
  - Research Site 10001-150, Los Angeles, California
  - Research Site 90001-005, Mission Viejo, California
  - Research Site 10001-043, Northridge, California
  - Research Site 10001-022, Northridge, California
  - Research Site 10001-033, Sacramento, California
  - Research Site 10001-105, San Ramon, California
  - Research Site 10001-008, Santa Rosa, California
  - Research Site 10001-153, Spring Valley, California
  - Research Site 90001-015, Stanford, California
  - Research Site 10001-044, Torrance, California
  - Research Site 90001-047, Boca Raton, Florida
  - Research Site 10001-084, Clearwater, Florida
  - Research Site 10001-155, Clearwater, Florida
  - Research Site 10001-099, Clearwater, Florida
  - Research Site 10001-127, Daytona Beach, Florida
  - Research Site 10001-119, Fleming Island, Florida
  - Research Site 10001-070, Fort Lauderdale, Florida
  - Research Site 10001-067, Hialeah, Florida
  - Research Site 10001-139, Jacksonville, Florida
  - Research Site 10001-039, Jacksonville, Florida
  - Research Site 10001-098, Jacksonville, Florida
  - Research Site 10001-081, Miami, Florida
  - Research Site 10001-140, Miami, Florida
  - Research Site 10001-142, Miami, Florida
  - Research Site 10001-030, Miami, Florida
  - Research Site 10001-116, Miami, Florida
  - Research Site 10001-080, Miami Springs, Florida
  - Research Site 10001-027, Pembroke Pines, Florida
  - Research Site 10001-115, Pembroke Pines, Florida
  - Research Site 10001-048, Pembroke Pines, Florida
  - Research Site 10001-147, Pembroke Pines, Florida
  - Research Site 10001-003, Pinellas Park, Florida
  - Research Site 10001-104, Ponte Vedra, Florida
  - Research Site 10001-090, Saint Augustine, Florida
  - Research Site 10001-123, Sarasota, Florida
  - Research Site 10001-102, St. Petersburg, Florida
  - Research Site 10001-143, Tampa, Florida
  - Research Site 10001-069, Atlanta, Georgia
  - Research Site 10001-137, Dunwoody, Georgia
  - Research Site 10001-092, Macon, Georgia
  - Research Site 10001-059, Arlington Heights, Illinois
  - Research Site 10001-158, Chicago, Illinois
  - Research Site 10001-036, Evanston, Illinois
  - Research Site 10001-082, Indianapolis, Indiana
  - Research Site 10001-040, Valparaiso, Indiana
  - Research Site 10001-074, West Des Moines, Iowa
  - Research Site 10001-028, Hutchinson, Kansas
  - Research Site 10001-125, Lexington, Kentucky
  - Research Site 10001-108, Lexington, Kentucky
  - Research Site 10001-107, Owensboro, Kentucky
  - Research Site 10001-144, Crowley, Louisiana
  - Research Site 10001-041, Lake Charles, Louisiana
  - Research Site 10001-101, Monroe, Louisiana
  - Research Site 90001-004, Boston, Massachusetts
  - Research Site 10001-024, Flint, Michigan
  - Research Site 10001-095, Grandville, Michigan
  - Research Site 10001-078, Sterling Heights, Michigan
  - Research Site 10001-034, Troy, Michigan
  - Research Site 10001-018, Edina, Minnesota
  - Research Site 90001-056, Saint Paul, Minnesota
  - Research Site 10001-156, St Louis, Missouri
  - Research Site 10001-007, St Louis, Missouri
  - Research Site 90001-012, Butte, Montana
  - Research Site 10001-053, Omaha, Nebraska
  - Research Site 10001-021, Omaha, Nebraska
  - Research Site 90001-112, Las Vegas, Nevada
  - Research Site 10001-124, Las Vegas, Nevada
  - Research Site 10001-060, Bridgewater, New Jersey
  - Research Site 90001-014, Summit, New Jersey
  - Research Site 10001-055, Warren Township, New Jersey
  - Research Site 10001-054, Albany, New York
  - Research Site 10001-122, Binghamton, New York
  - Research Site 10001-128, Endwell, New York
  - Research Site 10001-042, New Windsor, New York
  - Research Site 10001-129, Poughkeepsie, New York
  - Research Site 10001-110, Williamsville, New York
  - Research Site 10001-063, Cary, North Carolina
  - Research Site 10001-064, Greensboro, North Carolina
  - Research Site 10001-145, Mooresville, North Carolina
  - Research Site 10001-046, Shelby, North Carolina
  - Research Site 10001-016, Akron, Ohio
  - Research Site 10001-120, Cincinnati, Ohio
  - Research Site 90001-002, Cincinnati, Ohio
  - Research Site 10001-010, Cincinnati, Ohio
  - Research Site 10001-134, Cincinnati, Ohio
  - Research Site 10001-014, Columbus, Ohio
  - Research Site 10001-141, Dayton, Ohio
  - Research Site 10001-148, Marion, Ohio
  - Research Site 10001-109, Wyomissing, Pennsylvania
  - Research Site 10001-001, Anderson, South Carolina
  - Research Site 10001-006, Greer, South Carolina
  - Research Site 10001-075., Greer, South Carolina
  - Research Site 10001-111, Myrtle Beach, South Carolina
  - Research Site 10001-133, Pelzer, South Carolina
  - Research Site 10001-103, Rapid City, South Dakota
  - Research Site 10001-146, Athens, Tennessee
  - Research Site 10001-130, Kingsport, Tennessee
  - Research Site 10001-118, Knoxville, Tennessee
  - Research Site 10001-106, Knoxville, Tennessee
  - Research Site 10001-100, Amarillo, Texas
  - Research Site 10001-087, Austin, Texas
  - Research Site 10001-117, Austin, Texas
  - Research Site 10001-009, Dallas, Texas
  - Research Site 10001-068, Edinburg, Texas
  - Research Site 10001-031, Houston, Texas
  - Research Site 10001-088, Houston, Texas
  - Research Site 10001-091, Houston, Texas
  - Research Site 10001-061, Houston, Texas
  - Research Site 10001-032, Houston, Texas
  - Research Site 10001-057, New Braunfels, Texas
  - Research Site 10001-079, Round Rock, Texas
  - Research Site 10001-071, San Antonio, Texas
  - Research Site 10001-083, Schertz, Texas
  - Research Site 10001-149, Shavano Park, Texas
  - Research Site 10001-045, Tomball, Texas
  - Research Site 10001-005, Layton, Utah
  - Research Site 10001-002, Salt Lake City, Utah
  - Research Site 10001-052, Salt Lake City, Utah
  - Research Site 10001-093, Falls Church, Virginia
  - Research Site 10001-085, Manassas, Virginia
  - Research Site 10001-094, Midlothian, Virginia
  - Research Site 10001-023, Richmond, Virginia
  - Research Site 10001-029, Suffolk, Virginia
  - Research Site 10001-114, Tacoma, Washington
- Canada (3):
  - Research Site 90011-005, Chicoutimi, Quebec
  - Research Site 90011-001, Montreal, Quebec
  - Research Site 90011-002, Québec, Quebec
- Czechia (4):
  - Research Site 11420-002, Chomutov
  - Research Site 90420-001, Prague
  - Research Site 90420-006, Prague
  - Research Site 11420-003, Uherské Hradiště
- Denmark (6):
  - Research Site 90045-001, Aalborg, North Denmark
  - Research Site 90045-004, Esbjerg
  - Research Site 90045-003, Herning
  - Research Site 90045-006, Hvidovre
  - Research Site 90045-002, Roskilde
  - Research Site 90045-005, Viborg
- Germany (5):
  - Research Site 11049-006, Berlin
  - Research Site 11049-002, Bochum
  - Research Site 11049-003, Frankfurt
  - Research Site 11049-001, Heidelberg
  - Research Site 11049-007, Heidelberg
- Hungary (4):
  - Research Site 11036-001, Budapest
  - Research Site 11036-004, Debrecen
  - Research Site 11036-002, Hatvan
  - Research Site 11036-003, Zalaegerszeg
- Netherlands (5):
  - Research Site 90031-001, Amersfoort
  - Research Site 90031-003, Amsterdam
  - Research Site 90031-006, Goes
  - Research Site 90031-009, Hoorn
  - Research Site 90031-005, Utrecht
- Poland (18):
  - Research SIte 11048-016, Brzozowie
  - Research Site 11048-018, Bydgoszcz
  - Research Site 11048-011, Bydgoszcz
  - Research Site 11048-004, Gdansk
  - Research Site 11048-005, Gdynia
  - Research Site 11048-007, Katowice
  - Research SIte 11048-012, Katowice
  - Research Site 11048-003, Krakow
  - Research SIte 11048-014, Krakow
  - Research Site 11048-008, Lublin
  - Research Site 11048-001, Poznan
  - Research Site 11048-019, Ruda Śląska
  - Research SIte 11048-013, Rzeszów
  - Research SIte 11048-015, Tarnów
  - Research Site 11048-006, Warsaw
  - Research Site 11048-009, Warsaw
  - Research Site 11048-002, Wroclaw
  - Research Site 11048-010, Wroclaw
- South Africa (12):
  - Research Site 90027-008, Bellville, Cape Town
  - Research Site 90027-007, Lyttelton, Cape Town
  - Research Site 90027-003, Bloemfontein, Free State
  - Research Site 90027-010, Johannesburg, Gauteng
  - Research Site 11027-005, Kempton Park, Gauteng
  - Research Site 90027-006, Pretoria, Gauteng
  - Research Site 90027-009, Witbank, Gauteng
  - Research Site 90027-001, Cape Town, Western Cape
  - Research Site 11027-007, Kuils River, Western Cape
  - Research Site 11027-013, Paarl, Western Cape
  - Research Site 90027-004, Somerset West, Western Cape
  - Research Site 90027-005, Somerset West, Western Cape
- Spain (6):
  - Research Site 90034-004, Córdoba, Andalusia
  - Research Site 90034-002, Zaragoza, Aragon
  - Research Site 90034-005, Barcelona, Catalonia
  - Research Site 90034-006, Barcelona, Catalonia
  - Research Site 90034-001, Reus, Catalonia
  - Research Site 90034-003, A Coruña, Galicia
- Sweden (3):
  - Research Site 90046-002, Gothenburg
  - Research Site 90046-001, Stockholm
  - Research Site 90046-003, Stockholm
- Ukraine (8):
  - Research Site 11380-005, Cherkasy
  - Research Site 11380-008, Kharkiv
  - Research Site 11380-001, Kyiv
  - Research Site 11380-002, Kyiv
  - Research Site 11380-003, Kyiv
  - Research Site 11380-004, Kyiv
  - Research Site 11380-006, Uzhhorod
  - Research Site 11380-009, Zaporizhzhya
- United Kingdom (23):
  - Research Site 11044-028, Bollington, Cheshire
  - Research Site 11044-026, Bury
  - Research Site 11044-024, Cheadle Hulme
  - Research Site 11044-014, Chorley
  - Research Site 11044-012, Cornwell
  - Research Site 11044-010, Derby
  - Research Site 11044-006, Edgbaston
  - Research Site 11044-009, Exeter
  - Research Site 11044-001, Glasgow
  - Research Site 11044-008, Hexham
  - Research SIte 11044-020, Macclesfield
  - Research Site 11044-005, Manchester
  - Research Site 11044-025, Manchester
  - Research Site 11044-027, Manchester
  - Research Site 11044-029, Manchester
  - Research Site 11044-019, Plymouth
  - Research Site 11044-003, Reading
  - Research Site 11044-022, Sale
  - Research Site 11044-023, Sale
  - Research Site 11044-002, Stockton-on-Tees
  - Research Site 11044-021, Timperley
  - Research Site 11044-007, Wales
  - Research Site 11044-004, Waterloo

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Wright RS, Raal FJ, Koenig W, Landmesser U, Leiter LA, Vikarunnessa S, Lesogor A, Maheux P, Talloczy Z, Zang X, Schwartz GG, Ray KK. Inclisiran administration potently and durably lowers LDL-C over an extended-term follow-up: the ORION-8 trial. Cardiovasc Res. 2024 Oct 14;120(12):1400-1410. doi: 10.1093/cvr/cvae109. PMID 38753448
- [Derived] Warden BA, Duell PB. Inclisiran: A Novel Agent for Lowering Apolipoprotein B-containing Lipoproteins. J Cardiovasc Pharmacol. 2021 Aug 1;78(2):e157-e174. doi: 10.1097/FJC.0000000000001053. PMID 33990512

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 268 centers in 13 countries: United States(145), Canada(8), Czechia(4), Denmark(6), Germany(9), Hungary(4), Netherlands(12), Poland(18), South Africa(12), Spain(6), Sweden(3), Ukraine(8), United Kingdom(33)
Pre-assignment Details: Participants completed a qualifying Phase II lipid lowering trial [MDCO-PCS-16-01 (ORION-3)] or Phase III lipid-lowering ORION feeder study [MDCO-PCS-17-03 (ORION-9), MDCO-PCS-17-04 (ORION-10), or MDCO-PCS-17-08 (ORION-11) ] meaning the subject received the last dose of study drug and completed the final study visit per applicable protocol.
Groups:
- Phase III Inclisiran-Inclisiran: Subjects who received inclisiran (actual treatment) in studies ORION-9/ ORION-10/ORION-11
- Phase III Placebo-Inclisiran: subjects who received placebo (actual treatment) in ORION-9/ORION-10/ORION-11
- ORION-3 Rollover: Subjects rolling over from ORION-3 Phase II study
Period: Overall Study
Arm/Group | Phase III Inclisiran-Inclisiran | Phase III Placebo-Inclisiran | ORION-3 Rollover
Started (All enrolled participants) | 1513 | 1478 | 284
Safety Population (All ORION-3 rollover subjects who signed the informed consent to Study ORION-8, and all ORION-9/ORION-10/ORION-11 rollover subjects with at least one study drug administration in Study ORION-8) | 1512 (One patient discontinued before receiving the study treatment. Hence safety population has one less patient.) | 1478 | 284
Completed | 1246 | 1200 | 0
Not Completed | 267 | 278 | 284
Not completed — Sponsor's Administrative Decision | 0 | 0 | 272
Not completed — Death | 80 | 81 | 4
Not completed — Withdrew Consent | 77 | 78 | 2
Not completed — Lost to Follow-up | 47 | 52 | 1
Not completed — Adverse Event | 22 | 23 | 0
Not completed — Physician Decision | 7 | 4 | 2
Not completed — Initiation Of Protocol-Prohibited Approved PCSK9 Inhibitor | 0 | 0 | 1
Not completed — Other reasons | 34 | 40 | 2

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics are based on the safety population, as primary and secondary analysis are based on the safety population.
  The safety population consisted of all ORION-3 rollover subjects who signed the informed consent to Study ORION-8, and all ORION-9/ORION-10/ORION-11 rollover subjects with at least one study drug administration in Study ORION-8
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase III Inclisiran-Inclisiran | Phase III Placebo-Inclisiran | ORION-3 Rollover | Total
Number analyzed (Participants) | 1512 | 1478 | 284 | 3274
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (9.83) | 64.6 (9.82) | 67.7 (9.97) | 64.9 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 482 | 476 | 100 | 1058
  Male | 1030 | 1002 | 184 | 2216
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska Native | 3 | 2 | 2 | 7
  Asian | 17 | 7 | 3 | 27
  Black/African American | 103 | 78 | 7 | 188
  Native Hawaiian/Other Pacific Islander | 6 | 4 | 0 | 10
  White | 1383 | 1387 | 271 | 3041
  Missing | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving Global Lipid Targets for Their Level of ASCVD Risk
Description: The primary objective of the study is to evaluate the effect of inclisiran treatment on the proportion of subjects achieving prespecified LDL-C targets at end of study (EOS).
  Target is <70 mg/dL for atherosclerotic cardiovascular disease (ASCVD) subjects and <100 mg/dL for ASCVD risk equivalent subjects.
  Risk equivalent subjects are defined as either type 2 diabetes, familial hypercholesterolemia or a 10-year risk of a cardiovascular event ≥20% as assessed by the Framingham Risk Score or equivalent; without a medical history of coronary heart disease , cerebrovascular disease or peripheral artery disease.
Time Frame: From ORION-8 Day 1 to the end of study (up to 1080 days)
Population: Safety Population: All ORION-3 rollover subjects who signed the informed consent to Study ORION-8, and all ORION-9/ORION-10/ORION-11 rollover subjects with at least one study drug administration in Study. Only participants with valid LDL-C measurements at Day 1080/EOS were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Total: Total
Arm/Group | Phase III Inclisiran-Inclisiran | Phase III Placebo-Inclisiran | ORION-3 Rollover | Total
Number analyzed (Participants) | 1251 | 1204 | 276 | 2731
Percentage of participants
  % of subjects Who Attain Global Lipid Targets at Day 1080 / EOS | 78.18 [75.8 to 80.4] | 79.07 [76.7 to 81.3] | 76.81 [71.4 to 81.6] | 78.43 [76.8 to 80.0]
  % of ASCVD subjects Who Attain Global Lipid Targets of <70 mg/dL at Day 1080 / EOS: number analyzed (Participants) | 1036 | 993 | 176 | 2205
  % of ASCVD subjects Who Attain Global Lipid Targets of <70 mg/dL at Day 1080 / EOS | 79.34 [76.8 to 81.7] | 79.96 [77.4 to 82.4] | 76.70 [70.0 to 82.5] | 79.41 [77.7 to 81.1]
  % of ASCVD Risk Equivalent subjects Who Attain Global Lipid Targets of <100 mg/dL at Day 1080 / EOS: number analyzed (Participants) | 215 | 211 | 100 | 526
  % of ASCVD Risk Equivalent subjects Who Attain Global Lipid Targets of <100 mg/dL at Day 1080 / EOS | 72.56 [66.1 to 78.3] | 74.88 [68.6 to 80.5] | 77.00 [67.7 to 84.7] | 74.33 [70.4 to 78.0]

2. Primary Outcome: Incidence of Treatment-emergent Adverse Events (TEAEs)
Description: Safety assessments include adverse events and serious adverse events until the end of study.
  End of study visit occured at least 90 days following the last inclisiran dose once a decision was made to end the study (either by the subject, investigator or sponsor). For subjects prematurely and permanently discontinued from study treatment, who were not willing to return within the 90 day timeframe, the EOS visit was scheduled as soon as possible, or if decision to discontinue and not return was made at a specific visit, this visit became the EOS visit.
Time Frame: From ORION-8 Day 1 to the end of study (up to 1080 days)
Population: Safety Population: All ORION-3 rollover subjects who signed the informed consent to Study Orion-8, and all ORION-9/ORION-10/ORION-11 rollover subjects with at least one study drug administration in Study
Measure: Count of Participants; unit: Participants
Arm/Group | Phase III Inclisiran-Inclisiran | Phase III Placebo-Inclisiran | ORION-3 Rollover | Total
Number analyzed (Participants) | 1512 | 1478 | 284 | 3274
Participants
  Adverse events | 1197 | 1170 | 181 | 2548
  Adverse events :Treatment-related | 133 | 148 | 16 | 297
  SAEs | 464 | 482 | 43 | 989
  SAEs: Treatment-related | 2 | 2 | 1 | 5
  Fatal SAEs | 80 | 81 | 4 | 165
  Fatal SAEs: Treatment-related | 0 | 0 | 0 | 0

3. Secondary Outcome: Absolute Change in LDL-C From the Initial Feeder Study Baseline
Description: Absolute change from baseline in low density lipoprotein cholesterol (LDL-C) was calculated to evaluate the effect of inclisiran on LDL-C levels.
Time Frame: Feeder study baseline, ORION-8 baseline, Day 1080/EOS (ORION-8) (up to a maximum of 2340 days)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Phase III Inclisiran-Inclisiran | Phase III Placebo-Inclisiran | ORION-3 Rollover
Number analyzed (Participants) | 1512 | 1478 | 284
mg/dL
  ORION-8 Baseline | -55.21 [-56.9 to -53.5] | 0.46 [-1.4 to 2.3] | -61.58 [-66.4 to -56.8]
  Day 1080 / EOS: number analyzed (Participants) | 1251 | 1204 | 276
  Day 1080 / EOS | -55.81 [-58.0 to -53.6] | -54.70 [-56.9 to -52.5] | -64.31 [-69.0 to -59.7]

4. Secondary Outcome: Percentage Change in LDL-C From the Initial Feeder Study Baseline
Description: Percentage change from baseline in low density lipoprotein cholesterol (LDL-C) was calculated to evaluate the effect of inclisiran on LDL-C levels.
Time Frame: Feeder study baseline, ORION-8 baseline, Day 1080/EOS (ORION-8) (up to a maximum of 2340 days)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Percentage change in LDL-C
Arm/Group | Phase III Inclisiran-Inclisiran | Phase III Placebo-Inclisiran | ORION-3 Rollover
Number analyzed (Participants) | 1512 | 1478 | 284
Percentage change in LDL-C
  ORION-8 Baseline | -50.02 [-51.3 to -48.8] | 3.10 [1.4 to 4.9] | -48.22 [-51.2 to -45.2]
  Day 1080 / EOS: number analyzed (Participants) | 1251 | 1204 | 276
  Day 1080 / EOS | -48.96 [-50.5 to -47.4] | -49.69 [-51.3 to -48.0] | -49.95 [-52.6 to -47.3]

5. Secondary Outcome: Absolute Change From the Initial Feeder Study Baseline in Total Cholesterol, Triglycerides and HDL-C
Description: Absolute change from baseline in total cholesterol, triglycerides and high density lipoprotein cholesterol (HDL-C) was calculated to evaluate the effect of inclisiran on other lipids and lipoproteins.
Time Frame: Feeder study baseline, ORION-8 baseline, Day 1080/EOS (ORION-8) (up to a maximum of 2340 days)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Phase III Inclisiran-Inclisiran | Phase III Placebo-Inclisiran | ORION-3 Rollover
Number analyzed (Participants) | 1512 | 1478 | 284
mg/dL
  ORION-8 Baseline Total Cholesterol (TC) | -59.05 [-61.0 to -57.1] | -0.07 [-2.2 to 2.1] | -63.11 [-68.3 to -57.9]
  Day 1080 / EOS Total Cholesterol (TC): number analyzed (Participants) | 1251 | 1205 | 276
  Day 1080 / EOS Total Cholesterol (TC) | -58.48 [-61.0 to -55.9] | -57.08 [-59.6 to -54.6] | -65.43 [-70.5 to -60.3]
  ORION-8 Baseline Triglycerides | -21.50 [-25.1 to -17.9] | -5.74 [-9.5 to -2.0] | -14.43 [-23.7 to -5.1]
  Day 1080 / EOS Triglycerides: number analyzed (Participants) | 1251 | 1205 | 276
  Day 1080 / EOS Triglycerides | -19.58 [-23.7 to -15.4] | -22.12 [-26.3 to -17.9] | -21.32 [-30.3 to -12.4]
  ORION-8 Baseline HDL Cholesterol | 3.37 [2.9 to 3.9] | 0.59 [0.1 to 1.1] | 3.41 [2.2 to 4.6]
  Day 1080 / EOS HDL Cholesterol: number analyzed (Participants) | 1251 | 1205 | 276
  Day 1080 / EOS HDL Cholesterol | 3.60 [3.0 to 4.2] | 4.39 [3.8 to 5.0] | 5.27 [3.8 to 6.7]

6. Secondary Outcome: Percentage Change From the Initial Feeder Study Baseline in Total Cholesterol, Triglycerides and HDL-C
Description: Percentage change from baseline in total cholesterol (TC), triglycerides and high density lipoprotein cholesterol (HDL-C) was calculated to evaluate the effect of inclisiran on other lipids and lipoproteins.
Time Frame: Feeder study baseline, ORION-8 baseline, Day 1080/EOS (ORION-8) (up to a maximum of 2340 days)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Phase III Inclisiran-Inclisiran | Phase III Placebo-Inclisiran | ORION-3 Rollover
Number analyzed (Participants) | 1512 | 1478 | 284
Percentage change
  ORION-8 Baseline Total Cholesterol (TC) | -30.64 [-31.5 to -29.7] | 1.28 [0.1 to 2.4] | -29.49 [-31.6 to -27.4]
  Day 1080 / EOS Total Cholesterol (TC): number analyzed (Participants) | 1251 | 1205 | 276
  Day 1080 / EOS Total Cholesterol (TC) | -29.34 [-30.5 to -28.2] | -29.53 [-30.7 to -28.4] | -30.44 [-32.4 to -28.5]
  ORION-8 Baseline Triglycerides | -7.84 [-10.0 to -5.7] | 3.03 [0.8 to 5.2] | -0.20 [-7.6 to 7.2]
  Day 1080 / EOS Triglycerides: number analyzed (Participants) | 1251 | 1205 | 276
  Day 1080 / EOS Triglycerides | -3.90 [-6.5 to -1.3] | -6.85 [-9.2 to -4.5] | -3.18 [-9.2 to 2.8]
  ORION-8 Baseline HDL Cholesterol | 9.28 [8.2 to 10.4] | 3.48 [2.4 to 4.6] | 8.13 [5.7 to 10.5]
  Day 1080 / EOS HDL Cholesterol: number analyzed (Participants) | 1251 | 1205 | 276
  Day 1080 / EOS HDL Cholesterol | 9.91 [8.7 to 11.2] | 11.75 [10.3 to 13.2] | 12.16 [9.3 to 15.0]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the start of study in ORION-8 until end of study treatment plus 90 days post treatment, up to a maximum duration of 1080 days.
Description: Adverse Events are assessed in the safety population.
Arm/Group | Phase III Inclisiran-Inclisiran | Phase III Placebo-Inclisiran | ORION-3 Rollover | Total
All-Cause Mortality (participants affected / at risk) | 80/1512 | 81/1478 | 4/284 | 165/3274
Serious Adverse Events (participants affected / at risk) | 464/1512 | 482/1478 | 43/284 | 989/3274
Other Adverse Events (participants affected / at risk) | 1110/1512 | 1073/1478 | 169/284 | 2352/3274
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase III Inclisiran-Inclisiran (N=1512) | Phase III Placebo-Inclisiran (N=1478) | ORION-3 Rollover (N=284) | Total (N=3274)
Anaemia (Blood and lymphatic system disorders) | 3 | 4 | 0 | 7
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 3 | 3 | 0 | 6
Deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 3 | 0 | 5
Acute left ventricular failure (Cardiac disorders) | 2 | 0 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 17 | 24 | 3 | 44
Angina pectoris (Cardiac disorders) | 21 | 20 | 2 | 43
Angina unstable (Cardiac disorders) | 12 | 18 | 2 | 32
Aortic valve calcification (Cardiac disorders) | 0 | 1 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 3 | 3 | 0 | 6
Arrhythmic storm (Cardiac disorders) | 1 | 1 | 0 | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 2 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 17 | 15 | 3 | 35
Atrial flutter (Cardiac disorders) | 1 | 2 | 0 | 3
Atrioventricular block complete (Cardiac disorders) | 2 | 3 | 0 | 5
Atrioventricular block second degree (Cardiac disorders) | 1 | 1 | 0 | 2
Bradycardia (Cardiac disorders) | 2 | 4 | 0 | 6
Cardiac arrest (Cardiac disorders) | 3 | 6 | 0 | 9
Cardiac disorder (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 10 | 15 | 1 | 26
Cardiac failure acute (Cardiac disorders) | 4 | 3 | 0 | 7
Cardiac failure chronic (Cardiac disorders) | 3 | 3 | 0 | 6
Cardiac failure congestive (Cardiac disorders) | 15 | 13 | 1 | 29
Cardio-respiratory arrest (Cardiac disorders) | 2 | 2 | 0 | 4
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 3 | 0 | 0 | 3
Cardiorenal syndrome (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0 | 0 | 1
Chronic coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 1
Chronic left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 36 | 26 | 2 | 64
Coronary artery occlusion (Cardiac disorders) | 2 | 1 | 0 | 3
Coronary artery stenosis (Cardiac disorders) | 0 | 2 | 0 | 2
Diastolic dysfunction (Cardiac disorders) | 1 | 0 | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 1 | 0 | 2
Myocardial infarction (Cardiac disorders) | 12 | 19 | 2 | 33
Myocardial ischaemia (Cardiac disorders) | 7 | 8 | 0 | 15
Nodal arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 1
Prinzmetal angina (Cardiac disorders) | 1 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 2 | 0 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1 | 2
Supraventricular tachycardia (Cardiac disorders) | 1 | 1 | 0 | 2
Ventricular extrasystoles (Cardiac disorders) | 3 | 0 | 1 | 4
Ventricular fibrillation (Cardiac disorders) | 2 | 3 | 0 | 5
Ventricular hypokinesia (Cardiac disorders) | 1 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 4 | 6 | 0 | 10
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 1
Ear canal stenosis (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Otosclerosis (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 2 | 0 | 4
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Goitre (Endocrine disorders) | 0 | 1 | 0 | 1
Hyperparathyroidism primary (Endocrine disorders) | 1 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 1
Thyroiditis (Endocrine disorders) | 1 | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 1 | 0 | 2
Diplopia (Eye disorders) | 1 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 1 | 1 | 0 | 2
Retinal vein thrombosis (Eye disorders) | 0 | 1 | 0 | 1
Abdominal fat apron (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 2 | 0 | 8
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3 | 0 | 5
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 5 | 0 | 0 | 5
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 0 | 5
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastric fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastric volvulus (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 4 | 0 | 9
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 2 | 1 | 0 | 3
Intestinal atony (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1 | 0 | 3
Intestinal polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Oesophageal dysplasia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Oesophageal mucosal tear (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 4 | 1 | 0 | 5
Pancreatitis acute (Gastrointestinal disorders) | 4 | 1 | 0 | 5
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Proctitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pylorospasm (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Rectal prolapse (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Salivary duct obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 3 | 0 | 6
Small intestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Terminal ileitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 4 | 0 | 5
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3 | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Asthenia (General disorders) | 3 | 0 | 0 | 3
Chest discomfort (General disorders) | 0 | 1 | 0 | 1
Chest pain (General disorders) | 6 | 8 | 3 | 17
Death (General disorders) | 12 | 19 | 2 | 33
Exercise tolerance decreased (General disorders) | 1 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 1 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 10 | 10 | 0 | 20
Oedema peripheral (General disorders) | 1 | 1 | 0 | 2
Organ failure (General disorders) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Sudden cardiac death (General disorders) | 1 | 1 | 0 | 2
Swelling face (General disorders) | 1 | 0 | 0 | 1
Vascular stent occlusion (General disorders) | 1 | 0 | 0 | 1
Vascular stent stenosis (General disorders) | 1 | 1 | 0 | 2
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 4 | 1 | 7
Cholecystitis acute (Hepatobiliary disorders) | 3 | 6 | 0 | 9
Cholelithiasis (Hepatobiliary disorders) | 6 | 2 | 0 | 8
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Gallbladder rupture (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatic fibrosis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 1
Immunisation reaction (Immune system disorders) | 1 | 1 | 0 | 2
Sarcoidosis (Immune system disorders) | 1 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 2 | 0 | 0 | 2
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 1
Appendicitis (Infections and infestations) | 2 | 3 | 0 | 5
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 1 | 0 | 2
Bacteraemia (Infections and infestations) | 1 | 1 | 1 | 3
Bacterial colitis (Infections and infestations) | 0 | 1 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 2 | 0 | 3
COVID-19 (Infections and infestations) | 21 | 28 | 0 | 49
COVID-19 pneumonia (Infections and infestations) | 14 | 21 | 0 | 35
Cellulitis (Infections and infestations) | 7 | 7 | 1 | 15
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1 | 1
Device related infection (Infections and infestations) | 1 | 0 | 0 | 1
Diabetic foot infection (Infections and infestations) | 0 | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 2 | 0 | 3
Empyema (Infections and infestations) | 1 | 1 | 0 | 2
Endocarditis (Infections and infestations) | 1 | 1 | 0 | 2
Enterobacter infection (Infections and infestations) | 0 | 1 | 0 | 1
Enterobacter pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1
Epstein-Barr virus infection (Infections and infestations) | 0 | 1 | 0 | 1
Gangrene (Infections and infestations) | 2 | 2 | 0 | 4
Gastroenteritis (Infections and infestations) | 4 | 1 | 0 | 5
Gastroenteritis salmonella (Infections and infestations) | 1 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 1
Herpes zoster meningoencephalitis (Infections and infestations) | 1 | 0 | 0 | 1
Implant site infection (Infections and infestations) | 0 | 1 | 0 | 1
Infected bite (Infections and infestations) | 1 | 0 | 0 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0 | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 1 | 0 | 1
Labyrinthitis (Infections and infestations) | 1 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 4 | 0 | 5
Neuroborreliosis (Infections and infestations) | 1 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 2 | 4 | 0 | 6
Osteomyelitis chronic (Infections and infestations) | 1 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 16 | 17 | 2 | 35
Pneumonia bacterial (Infections and infestations) | 2 | 0 | 0 | 2
Pneumonia viral (Infections and infestations) | 1 | 1 | 0 | 2
Post procedural infection (Infections and infestations) | 0 | 0 | 1 | 1
Post-acute COVID-19 syndrome (Infections and infestations) | 1 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 1
Pyelitis (Infections and infestations) | 0 | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 1 | 0 | 2
Sepsis (Infections and infestations) | 4 | 8 | 3 | 15
Septic shock (Infections and infestations) | 1 | 5 | 0 | 6
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 2
Skin infection (Infections and infestations) | 1 | 0 | 0 | 1
Streptococcal urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 9 | 5 | 0 | 14
Urosepsis (Infections and infestations) | 3 | 0 | 1 | 4
Viraemia (Infections and infestations) | 1 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 1
Wound infection (Infections and infestations) | 2 | 2 | 0 | 4
Wound sepsis (Infections and infestations) | 0 | 2 | 0 | 2
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 4 | 0 | 6
Aortic restenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 6 | 0 | 0 | 6
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 3
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 3
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 3
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Rib fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Stomal hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 3
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 3
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Vascular access site haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Anticoagulation drug level above therapeutic (Investigations) | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 1
Myocardial necrosis marker increased (Investigations) | 0 | 1 | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 1 | 0 | 1
Troponin T increased (Investigations) | 0 | 1 | 0 | 1
Troponin increased (Investigations) | 0 | 1 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 1 | 0 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 2 | 0 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 4 | 0 | 0 | 4
Gout (Metabolism and nutrition disorders) | 1 | 2 | 0 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 3
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 3 | 0 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 3
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 0 | 7
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 0 | 0 | 8
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 4
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 3
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 5 | 3 | 1 | 9
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 16 | 20 | 0 | 36
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 4
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 3
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 3
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 4
Spinal synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Anaplastic thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 3
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2 | 1 | 8
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5 | 1 | 8
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Brenner tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 2
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5 | 0 | 7
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 2
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 2
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Laryngeal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 2
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 4 | 0 | 11
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 2
Malignant glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Malignant mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 0 | 5
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 3
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Non-Hodgkin's lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 2
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 3
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 4
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 2
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 7 | 0 | 15
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Sarcoma uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1 | 5
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0 | 4
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 0 | 5
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Triple negative breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 1
Basal ganglia haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 1
Bell's palsy (Nervous system disorders) | 1 | 1 | 0 | 2
Carotid arteriosclerosis (Nervous system disorders) | 0 | 1 | 0 | 1
Carotid artery disease (Nervous system disorders) | 1 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 2 | 2 | 0 | 4
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 1 | 1
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 1 | 1 | 3
Cerebral infarction (Nervous system disorders) | 2 | 2 | 0 | 4
Cerebral ischaemia (Nervous system disorders) | 1 | 1 | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 8 | 4 | 2 | 14
Cerebrovascular disorder (Nervous system disorders) | 1 | 0 | 0 | 1
Cervical cord compression (Nervous system disorders) | 0 | 1 | 0 | 1
Cortical laminar necrosis (Nervous system disorders) | 0 | 1 | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 2 | 0 | 4
Embolic stroke (Nervous system disorders) | 1 | 1 | 0 | 2
Encephalopathy (Nervous system disorders) | 3 | 1 | 0 | 4
Epilepsy (Nervous system disorders) | 2 | 0 | 0 | 2
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 1
Intracranial mass (Nervous system disorders) | 1 | 0 | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 16 | 10 | 0 | 26
Lacunar infarction (Nervous system disorders) | 2 | 1 | 0 | 3
Lacunar stroke (Nervous system disorders) | 0 | 2 | 0 | 2
Loss of consciousness (Nervous system disorders) | 4 | 0 | 0 | 4
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 1
Metabolic encephalopathy (Nervous system disorders) | 2 | 0 | 0 | 2
Migraine (Nervous system disorders) | 2 | 0 | 0 | 2
Myelopathy (Nervous system disorders) | 0 | 1 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1 | 0 | 1
Paralysis (Nervous system disorders) | 0 | 1 | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 1
Presyncope (Nervous system disorders) | 3 | 1 | 0 | 4
Sciatica (Nervous system disorders) | 1 | 1 | 0 | 2
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 1 | 0 | 3
Syncope (Nervous system disorders) | 11 | 6 | 1 | 18
Thalamus haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 5 | 7 | 1 | 13
Vascular encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 1
Vasogenic cerebral oedema (Nervous system disorders) | 1 | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 1 | 0 | 1
Device loosening (Product Issues) | 0 | 1 | 0 | 1
Device malfunction (Product Issues) | 1 | 1 | 0 | 2
Device occlusion (Product Issues) | 0 | 1 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 1 | 0 | 2
Confusional state (Psychiatric disorders) | 1 | 3 | 0 | 4
Conversion disorder (Psychiatric disorders) | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 0 | 2
Generalised anxiety disorder (Psychiatric disorders) | 1 | 0 | 0 | 1
Major depression (Psychiatric disorders) | 2 | 0 | 0 | 2
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 16 | 12 | 1 | 29
Chronic kidney disease (Renal and urinary disorders) | 2 | 2 | 0 | 4
End stage renal disease (Renal and urinary disorders) | 0 | 1 | 0 | 1
Glomerulonephritis chronic (Renal and urinary disorders) | 0 | 1 | 0 | 1
Glomerulonephritis membranous (Renal and urinary disorders) | 1 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 4 | 0 | 0 | 4
Hydronephrosis (Renal and urinary disorders) | 1 | 2 | 0 | 3
Nephrolithiasis (Renal and urinary disorders) | 2 | 4 | 0 | 6
Neurogenic bladder (Renal and urinary disorders) | 1 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 3 | 5 | 0 | 8
Renal haemorrhage (Renal and urinary disorders) | 0 | 2 | 0 | 2
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 1
Renal mass (Renal and urinary disorders) | 0 | 1 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 2 | 2 | 0 | 4
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 3 | 1 | 0 | 4
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 7 | 2 | 0 | 9
Breast necrosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Perineal fistula (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 2 | 0 | 0 | 2
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 | 17 | 2 | 28
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 0 | 17
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 8 | 2 | 16
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 5
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 4
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 3
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 0 | 14
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 3
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 6
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Reactive perforating collagenosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Aneurysm (Vascular disorders) | 1 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 5 | 7 | 0 | 12
Aortic dissection (Vascular disorders) | 0 | 1 | 1 | 2
Aortic occlusion (Vascular disorders) | 0 | 0 | 1 | 1
Aortic stenosis (Vascular disorders) | 3 | 6 | 0 | 9
Arterial stenosis (Vascular disorders) | 0 | 1 | 0 | 1
Arteriosclerosis (Vascular disorders) | 3 | 0 | 0 | 3
Circulatory collapse (Vascular disorders) | 0 | 2 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 2 | 1 | 0 | 3
Embolism venous (Vascular disorders) | 1 | 0 | 0 | 1
Essential hypertension (Vascular disorders) | 1 | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 0 | 0 | 1
Granulomatosis with polyangiitis (Vascular disorders) | 0 | 1 | 0 | 1
Haematoma (Vascular disorders) | 1 | 1 | 0 | 2
Hypertension (Vascular disorders) | 3 | 2 | 1 | 6
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 1
Hypertensive emergency (Vascular disorders) | 1 | 0 | 0 | 1
Hypertensive urgency (Vascular disorders) | 1 | 2 | 0 | 3
Hypotension (Vascular disorders) | 4 | 1 | 1 | 6
Intermittent claudication (Vascular disorders) | 2 | 0 | 0 | 2
Labile hypertension (Vascular disorders) | 0 | 1 | 0 | 1
Leriche syndrome (Vascular disorders) | 0 | 1 | 0 | 1
Penetrating aortic ulcer (Vascular disorders) | 1 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 5 | 8 | 0 | 13
Peripheral artery aneurysm (Vascular disorders) | 0 | 1 | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 3 | 1 | 0 | 4
Peripheral artery stenosis (Vascular disorders) | 1 | 0 | 0 | 1
Peripheral embolism (Vascular disorders) | 0 | 1 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 3 | 0 | 3
Peripheral vascular disorder (Vascular disorders) | 1 | 2 | 0 | 3
Varicose vein (Vascular disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase III Inclisiran-Inclisiran (N=1512) | Phase III Placebo-Inclisiran (N=1478) | ORION-3 Rollover (N=284) | Total (N=3274)
Anaemia (Blood and lymphatic system disorders) | 45 | 33 | 2 | 80
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 3 | 0 | 4
Anaemia megaloblastic (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2
Bone marrow oedema (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Cytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 2
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 10 | 4 | 0 | 14
Leukocytosis (Blood and lymphatic system disorders) | 8 | 4 | 0 | 12
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Lymph node fibrosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 3 | 1 | 6
Macrocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 3 | 5 | 1 | 9
Monoclonal B-cell lymphocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 0 | 4
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Normocytic anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 3
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Polycythaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 2
Splenomegaly (Blood and lymphatic system disorders) | 1 | 2 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 8 | 0 | 8
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 2
Angina pectoris (Cardiac disorders) | 24 | 32 | 2 | 58
Angina unstable (Cardiac disorders) | 4 | 3 | 0 | 7
Aortic valve incompetence (Cardiac disorders) | 4 | 4 | 0 | 8
Aortic valve sclerosis (Cardiac disorders) | 1 | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 2 | 5 | 0 | 7
Arrhythmia (Cardiac disorders) | 3 | 3 | 0 | 6
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 1 | 0 | 2
Atrial enlargement (Cardiac disorders) | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 40 | 36 | 4 | 80
Atrial flutter (Cardiac disorders) | 2 | 1 | 0 | 3
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Atrial thrombosis (Cardiac disorders) | 1 | 0 | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 3 | 3 | 0 | 6
Atrioventricular block second degree (Cardiac disorders) | 1 | 1 | 0 | 2
Bradycardia (Cardiac disorders) | 12 | 13 | 1 | 26
Bundle branch block (Cardiac disorders) | 1 | 0 | 0 | 1
Bundle branch block left (Cardiac disorders) | 1 | 2 | 0 | 3
Bundle branch block right (Cardiac disorders) | 1 | 2 | 0 | 3
Cardiac amyloidosis (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac aneurysm (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 15 | 19 | 0 | 34
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 3 | 1 | 0 | 4
Cardiac failure congestive (Cardiac disorders) | 15 | 11 | 0 | 26
Cardiac flutter (Cardiac disorders) | 1 | 1 | 0 | 2
Cardiac hypertrophy (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac perfusion defect (Cardiac disorders) | 1 | 1 | 0 | 2
Cardiac sarcoidosis (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac valve disease (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 2 | 0 | 0 | 2
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiomegaly (Cardiac disorders) | 3 | 1 | 0 | 4
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiorenal syndrome (Cardiac disorders) | 1 | 1 | 0 | 2
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 0 | 1
Chronic left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 1
Chronotropic incompetence (Cardiac disorders) | 0 | 1 | 0 | 1
Conduction disorder (Cardiac disorders) | 1 | 1 | 0 | 2
Congestive cardiomyopathy (Cardiac disorders) | 1 | 1 | 0 | 2
Coronary artery disease (Cardiac disorders) | 17 | 24 | 0 | 41
Coronary artery occlusion (Cardiac disorders) | 3 | 0 | 0 | 3
Coronary artery stenosis (Cardiac disorders) | 2 | 2 | 0 | 4
Diastolic dysfunction (Cardiac disorders) | 1 | 4 | 0 | 5
Dressler's syndrome (Cardiac disorders) | 0 | 1 | 0 | 1
Extrasystoles (Cardiac disorders) | 1 | 1 | 0 | 2
Heart valve incompetence (Cardiac disorders) | 2 | 0 | 0 | 2
Hypertensive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 1 | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 4 | 0 | 5
Left atrial enlargement (Cardiac disorders) | 0 | 1 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 3 | 4 | 0 | 7
Left ventricular enlargement (Cardiac disorders) | 1 | 0 | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 2 | 1 | 4
Left ventricular hypertrophy (Cardiac disorders) | 4 | 1 | 0 | 5
Mitral valve calcification (Cardiac disorders) | 1 | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 11 | 7 | 1 | 19
Mitral valve prolapse (Cardiac disorders) | 1 | 0 | 0 | 1
Mitral valve stenosis (Cardiac disorders) | 2 | 0 | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 4 | 5 | 0 | 9
Palpitations (Cardiac disorders) | 21 | 8 | 1 | 30
Pericardial effusion (Cardiac disorders) | 3 | 0 | 0 | 3
Pericarditis (Cardiac disorders) | 2 | 0 | 0 | 2
Prinzmetal angina (Cardiac disorders) | 0 | 1 | 0 | 1
Pulmonary valve incompetence (Cardiac disorders) | 2 | 1 | 0 | 3
Right atrial dilatation (Cardiac disorders) | 1 | 0 | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 0 | 2 | 1 | 3
Sinus bradycardia (Cardiac disorders) | 3 | 4 | 0 | 7
Sinus node dysfunction (Cardiac disorders) | 4 | 4 | 0 | 8
Sinus tachycardia (Cardiac disorders) | 3 | 3 | 0 | 6
Supraventricular extrasystoles (Cardiac disorders) | 4 | 1 | 0 | 5
Supraventricular tachycardia (Cardiac disorders) | 2 | 8 | 0 | 10
Systolic dysfunction (Cardiac disorders) | 0 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 7 | 6 | 1 | 14
Tachycardia paroxysmal (Cardiac disorders) | 1 | 0 | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 6 | 4 | 1 | 11
Ventricular arrhythmia (Cardiac disorders) | 0 | 2 | 0 | 2
Ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 9 | 3 | 1 | 13
Ventricular tachycardia (Cardiac disorders) | 5 | 9 | 0 | 14
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 1
Apolipoprotein E e4 gene carrier (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 1
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 1
Genetic polymorphism (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 2 | 0 | 2
Phimosis (Congenital, familial and genetic disorders) | 0 | 1 | 1 | 2
SF3B1 gene mutation (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 3 | 5 | 0 | 8
Conductive deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Deafness (Ear and labyrinth disorders) | 4 | 1 | 1 | 6
Deafness bilateral (Ear and labyrinth disorders) | 1 | 1 | 0 | 2
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 3 | 0 | 3
Deafness unilateral (Ear and labyrinth disorders) | 2 | 2 | 0 | 4
Ear canal stenosis (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 9 | 3 | 0 | 12
Ear pruritus (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 | 1 | 0 | 2
Excessive cerumen production (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Haematotympanum (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 3 | 1 | 4
Mastoid disorder (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 1 | 1 | 0 | 2
Otolithiasis (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 3 | 10 | 0 | 13
Vertigo (Ear and labyrinth disorders) | 15 | 14 | 4 | 33
Vertigo positional (Ear and labyrinth disorders) | 4 | 0 | 0 | 4
Adrenal mass (Endocrine disorders) | 1 | 1 | 0 | 2
Autoimmune thyroiditis (Endocrine disorders) | 1 | 4 | 0 | 5
Goitre (Endocrine disorders) | 2 | 4 | 0 | 6
Hyperparathyroidism (Endocrine disorders) | 1 | 3 | 0 | 4
Hyperparathyroidism primary (Endocrine disorders) | 1 | 0 | 0 | 1
Hyperprolactinaemia (Endocrine disorders) | 1 | 1 | 0 | 2
Hyperthyroidism (Endocrine disorders) | 6 | 5 | 0 | 11
Hypogonadism (Endocrine disorders) | 1 | 1 | 0 | 2
Hypothyroidism (Endocrine disorders) | 10 | 10 | 2 | 22
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1 | 0 | 1
Thyroid calcification (Endocrine disorders) | 0 | 1 | 0 | 1
Thyroid mass (Endocrine disorders) | 2 | 1 | 0 | 3
Age-related macular degeneration (Eye disorders) | 1 | 1 | 0 | 2
Amaurosis fugax (Eye disorders) | 1 | 0 | 0 | 1
Blepharitis (Eye disorders) | 2 | 0 | 0 | 2
Blepharospasm (Eye disorders) | 0 | 1 | 0 | 1
Blindness (Eye disorders) | 0 | 0 | 1 | 1
Cataract (Eye disorders) | 40 | 23 | 5 | 68
Chalazion (Eye disorders) | 0 | 2 | 0 | 2
Choroidal neovascularisation (Eye disorders) | 1 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 2 | 2 | 0 | 4
Conjunctivitis allergic (Eye disorders) | 2 | 1 | 0 | 3
Corneal degeneration (Eye disorders) | 1 | 0 | 0 | 1
Corneal erosion (Eye disorders) | 1 | 0 | 0 | 1
Dermatochalasis (Eye disorders) | 0 | 1 | 0 | 1
Diabetic retinopathy (Eye disorders) | 1 | 3 | 4 | 8
Diplopia (Eye disorders) | 2 | 1 | 0 | 3
Dry eye (Eye disorders) | 3 | 4 | 0 | 7
Ectropion (Eye disorders) | 0 | 1 | 1 | 2
Epiretinal membrane (Eye disorders) | 1 | 0 | 0 | 1
Exfoliation syndrome (Eye disorders) | 1 | 0 | 0 | 1
Eye discharge (Eye disorders) | 0 | 1 | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 1 | 0 | 1
Eye pain (Eye disorders) | 0 | 1 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 1
Eye swelling (Eye disorders) | 0 | 1 | 0 | 1
Eyelid cyst (Eye disorders) | 1 | 0 | 0 | 1
Eyelid ptosis (Eye disorders) | 1 | 1 | 0 | 2
Glaucoma (Eye disorders) | 5 | 7 | 1 | 13
Iridocyclitis (Eye disorders) | 0 | 0 | 1 | 1
Iritis (Eye disorders) | 1 | 0 | 0 | 1
Keratitis (Eye disorders) | 1 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 0 | 1 | 2
Macular degeneration (Eye disorders) | 7 | 1 | 1 | 9
Macular oedema (Eye disorders) | 0 | 2 | 0 | 2
Neovascular age-related macular degeneration (Eye disorders) | 0 | 1 | 0 | 1
Non-proliferative retinopathy (Eye disorders) | 0 | 1 | 0 | 1
Ocular hypertension (Eye disorders) | 0 | 0 | 1 | 1
Periorbital swelling (Eye disorders) | 0 | 1 | 0 | 1
Posterior capsule opacification (Eye disorders) | 0 | 1 | 0 | 1
Retinal artery embolism (Eye disorders) | 1 | 0 | 0 | 1
Retinal artery occlusion (Eye disorders) | 1 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 2 | 1 | 1 | 4
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0 | 1
Retinal ischaemia (Eye disorders) | 1 | 0 | 0 | 1
Retinal vascular thrombosis (Eye disorders) | 0 | 0 | 1 | 1
Retinal vein occlusion (Eye disorders) | 0 | 1 | 0 | 1
Retinopathy (Eye disorders) | 0 | 1 | 1 | 2
Retinopathy hypertensive (Eye disorders) | 1 | 0 | 0 | 1
Swelling of eyelid (Eye disorders) | 1 | 0 | 0 | 1
Ulcerative keratitis (Eye disorders) | 1 | 0 | 0 | 1
Vision blurred (Eye disorders) | 3 | 4 | 1 | 8
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 1
Visual impairment (Eye disorders) | 5 | 4 | 1 | 10
Vitreous detachment (Eye disorders) | 1 | 1 | 1 | 3
Vitreous floaters (Eye disorders) | 3 | 1 | 0 | 4
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0 | 1
Vitreous opacities (Eye disorders) | 1 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 7 | 1 | 8
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Abdominal hernia (Gastrointestinal disorders) | 2 | 1 | 1 | 4
Abdominal mass (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 15 | 16 | 3 | 34
Abdominal pain lower (Gastrointestinal disorders) | 3 | 2 | 1 | 6
Abdominal pain upper (Gastrointestinal disorders) | 6 | 11 | 3 | 20
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Acquired oesophageal web (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Anal prolapse (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Anal skin tags (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 2 | 1 | 4
Change of bowel habit (Gastrointestinal disorders) | 2 | 1 | 0 | 3
Chronic gastritis (Gastrointestinal disorders) | 2 | 3 | 0 | 5
Colitis (Gastrointestinal disorders) | 2 | 1 | 0 | 3
Colitis microscopic (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Colitis ulcerative (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 22 | 25 | 2 | 49
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Defaecation disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 5 | 4 | 0 | 9
Diarrhoea (Gastrointestinal disorders) | 41 | 31 | 4 | 76
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Diverticulitis oesophageal (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 5 | 4 | 0 | 9
Diverticulum intestinal (Gastrointestinal disorders) | 6 | 10 | 0 | 16
Dry mouth (Gastrointestinal disorders) | 4 | 0 | 0 | 4
Duodenal polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 2 | 2 | 0 | 4
Duodenitis (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 8 | 9 | 1 | 18
Dysphagia (Gastrointestinal disorders) | 11 | 5 | 1 | 17
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Eosinophilic oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 3 | 0 | 3
Erosive duodenitis (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Eructation (Gastrointestinal disorders) | 1 | 3 | 0 | 4
Faeces discoloured (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Faeces soft (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 4 | 7 | 0 | 11
Food poisoning (Gastrointestinal disorders) | 2 | 2 | 0 | 4
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastric disorder (Gastrointestinal disorders) | 1 | 2 | 1 | 4
Gastric mucosa erythema (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Gastritis (Gastrointestinal disorders) | 12 | 13 | 3 | 28
Gastritis erosive (Gastrointestinal disorders) | 3 | 3 | 0 | 6
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 16 | 23 | 5 | 44
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 4 | 3 | 0 | 7
Haemorrhoids (Gastrointestinal disorders) | 9 | 10 | 0 | 19
Hiatus hernia (Gastrointestinal disorders) | 7 | 10 | 2 | 19
Ileus (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 5 | 7 | 1 | 13
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Intestinal polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 2 | 2 | 1 | 5
Large intestine polyp (Gastrointestinal disorders) | 10 | 7 | 0 | 17
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 23 | 17 | 1 | 41
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 5 | 3 | 0 | 8
Pancreatic cyst (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Pancreatic duct dilatation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pancreatic failure (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Pancreatic steatosis (Gastrointestinal disorders) | 3 | 3 | 0 | 6
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 1 | 2 | 0 | 3
Peritoneal adhesions (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Proctitis (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Rectal discharge (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 3 | 2 | 7
Rectal polyp (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Rectal prolapse (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Regurgitation (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Salivary gland mass (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 2 | 0 | 4
Tongue cyst (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Toothache (Gastrointestinal disorders) | 2 | 3 | 0 | 5
Umbilical hernia (Gastrointestinal disorders) | 5 | 5 | 0 | 10
Vomiting (Gastrointestinal disorders) | 16 | 9 | 3 | 28
Adverse drug reaction (General disorders) | 1 | 3 | 1 | 5
Application site rash (General disorders) | 1 | 0 | 0 | 1
Asthenia (General disorders) | 12 | 8 | 0 | 20
Calcinosis (General disorders) | 1 | 0 | 0 | 1
Chest discomfort (General disorders) | 8 | 5 | 3 | 16
Chest pain (General disorders) | 16 | 15 | 5 | 36
Chills (General disorders) | 2 | 1 | 0 | 3
Crepitations (General disorders) | 1 | 0 | 0 | 1
Cyst (General disorders) | 2 | 0 | 0 | 2
Drug intolerance (General disorders) | 2 | 0 | 0 | 2
Exercise tolerance decreased (General disorders) | 6 | 2 | 0 | 8
Eye complication associated with device (General disorders) | 1 | 0 | 0 | 1
Facial pain (General disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 27 | 22 | 4 | 53
Feeling abnormal (General disorders) | 0 | 1 | 0 | 1
Gait disturbance (General disorders) | 2 | 4 | 1 | 7
Generalised oedema (General disorders) | 0 | 1 | 0 | 1
Hernia (General disorders) | 0 | 2 | 0 | 2
Inflammation (General disorders) | 1 | 1 | 0 | 2
Influenza like illness (General disorders) | 10 | 5 | 2 | 17
Injection site bruising (General disorders) | 3 | 3 | 0 | 6
Injection site eczema (General disorders) | 0 | 1 | 0 | 1
Injection site erythema (General disorders) | 10 | 12 | 2 | 24
Injection site hypersensitivity (General disorders) | 0 | 1 | 0 | 1
Injection site induration (General disorders) | 0 | 1 | 0 | 1
Injection site oedema (General disorders) | 0 | 1 | 0 | 1
Injection site pain (General disorders) | 22 | 17 | 0 | 39
Injection site paraesthesia (General disorders) | 1 | 6 | 0 | 7
Injection site pruritus (General disorders) | 2 | 4 | 0 | 6
Injection site rash (General disorders) | 9 | 7 | 0 | 16
Injection site reaction (General disorders) | 42 | 49 | 2 | 93
Injection site vesicles (General disorders) | 0 | 1 | 0 | 1
Injury associated with device (General disorders) | 0 | 1 | 0 | 1
Malaise (General disorders) | 0 | 2 | 0 | 2
Mass (General disorders) | 1 | 0 | 1 | 2
Mucosal inflammation (General disorders) | 0 | 2 | 0 | 2
Nodule (General disorders) | 2 | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 10 | 11 | 1 | 22
Oedema (General disorders) | 3 | 3 | 3 | 9
Oedema peripheral (General disorders) | 29 | 20 | 2 | 51
Pain (General disorders) | 7 | 5 | 1 | 13
Peripheral swelling (General disorders) | 13 | 14 | 0 | 27
Physical deconditioning (General disorders) | 0 | 1 | 0 | 1
Polyp (General disorders) | 1 | 0 | 1 | 2
Pyrexia (General disorders) | 8 | 13 | 0 | 21
Sensation of foreign body (General disorders) | 1 | 0 | 0 | 1
Swelling face (General disorders) | 2 | 0 | 0 | 2
Vessel puncture site bruise (General disorders) | 0 | 1 | 0 | 1
Vessel puncture site haemorrhage (General disorders) | 0 | 1 | 0 | 1
Alcoholic liver disease (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Biliary dilatation (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 3 | 0 | 4
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 1 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 11 | 16 | 1 | 28
Gallbladder polyp (Hepatobiliary disorders) | 0 | 3 | 0 | 3
Hepatic calcification (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 1 | 0 | 2
Hepatic cyst (Hepatobiliary disorders) | 0 | 6 | 0 | 6
Hepatic fibrosis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2 | 0 | 2
Hepatic haematoma (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatic lesion (Hepatobiliary disorders) | 1 | 2 | 0 | 3
Hepatic steatosis (Hepatobiliary disorders) | 17 | 17 | 4 | 38
Hepatomegaly (Hepatobiliary disorders) | 3 | 1 | 0 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 4 | 0 | 7
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 2 | 0 | 2
Liver injury (Hepatobiliary disorders) | 2 | 1 | 0 | 3
Non-alcoholic fatty liver (Hepatobiliary disorders) | 1 | 2 | 1 | 4
Allergy to arthropod bite (Immune system disorders) | 1 | 0 | 0 | 1
Allergy to arthropod sting (Immune system disorders) | 1 | 1 | 0 | 2
Contrast media allergy (Immune system disorders) | 1 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 3 | 3 | 1 | 7
Dust allergy (Immune system disorders) | 0 | 1 | 0 | 1
Food allergy (Immune system disorders) | 1 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 3 | 0 | 3
Immunisation reaction (Immune system disorders) | 5 | 7 | 1 | 13
Sarcoidosis (Immune system disorders) | 1 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 9 | 16 | 1 | 26
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 1
Abscess (Infections and infestations) | 1 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 3 | 2 | 0 | 5
Abscess of eyelid (Infections and infestations) | 1 | 0 | 0 | 1
Acarodermatitis (Infections and infestations) | 2 | 0 | 0 | 2
Acute sinusitis (Infections and infestations) | 10 | 7 | 0 | 17
Appendicitis (Infections and infestations) | 0 | 2 | 0 | 2
Arthritis infective (Infections and infestations) | 0 | 1 | 0 | 1
Aspergillus infection (Infections and infestations) | 1 | 0 | 0 | 1
Asymptomatic COVID-19 (Infections and infestations) | 4 | 1 | 0 | 5
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 1
Bacterial vaginosis (Infections and infestations) | 2 | 0 | 0 | 2
Bartholinitis (Infections and infestations) | 1 | 0 | 0 | 1
Blister infected (Infections and infestations) | 1 | 0 | 0 | 1
Body tinea (Infections and infestations) | 1 | 1 | 0 | 2
Borrelia infection (Infections and infestations) | 1 | 1 | 0 | 2
Breast cellulitis (Infections and infestations) | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 32 | 27 | 1 | 60
Bronchitis viral (Infections and infestations) | 1 | 0 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 178 | 176 | 52 | 406
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Candida infection (Infections and infestations) | 2 | 1 | 0 | 3
Cellulitis (Infections and infestations) | 20 | 20 | 3 | 43
Chronic sinusitis (Infections and infestations) | 2 | 5 | 0 | 7
Conjunctivitis (Infections and infestations) | 4 | 2 | 0 | 6
Conjunctivitis bacterial (Infections and infestations) | 1 | 1 | 0 | 2
Coronavirus infection (Infections and infestations) | 5 | 5 | 4 | 14
Cystitis (Infections and infestations) | 6 | 6 | 1 | 13
Dacryocystitis (Infections and infestations) | 0 | 1 | 0 | 1
Dermatophytosis of nail (Infections and infestations) | 1 | 1 | 0 | 2
Device related infection (Infections and infestations) | 0 | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 2 | 7 | 2 | 11
Ear infection (Infections and infestations) | 5 | 10 | 1 | 16
Eczema infected (Infections and infestations) | 2 | 0 | 0 | 2
Epididymitis (Infections and infestations) | 1 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 1
Erythema migrans (Infections and infestations) | 0 | 1 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
External ear cellulitis (Infections and infestations) | 0 | 1 | 0 | 1
Eye infection (Infections and infestations) | 0 | 1 | 0 | 1
Eye infection viral (Infections and infestations) | 1 | 0 | 0 | 1
Eyelid infection (Infections and infestations) | 1 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 3 | 0 | 0 | 3
Fungal foot infection (Infections and infestations) | 1 | 1 | 0 | 2
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 1
Fungal skin infection (Infections and infestations) | 0 | 1 | 1 | 2
Furuncle (Infections and infestations) | 0 | 2 | 0 | 2
Gangrene (Infections and infestations) | 1 | 1 | 1 | 3
Gastroenteritis (Infections and infestations) | 14 | 13 | 0 | 27
Gastroenteritis clostridial (Infections and infestations) | 1 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 2 | 6 | 0 | 8
Gastrointestinal viral infection (Infections and infestations) | 0 | 1 | 0 | 1
Genital candidiasis (Infections and infestations) | 0 | 0 | 1 | 1
Genital herpes (Infections and infestations) | 1 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 1 | 3 | 1 | 5
Groin abscess (Infections and infestations) | 3 | 0 | 0 | 3
Gynaecological chlamydia infection (Infections and infestations) | 1 | 0 | 0 | 1
Helicobacter gastritis (Infections and infestations) | 3 | 1 | 0 | 4
Helicobacter infection (Infections and infestations) | 0 | 5 | 1 | 6
Herpes dermatitis (Infections and infestations) | 0 | 1 | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0 | 1 | 2
Herpes virus infection (Infections and infestations) | 1 | 2 | 0 | 3
Herpes zoster (Infections and infestations) | 16 | 9 | 0 | 25
Herpes zoster infection neurological (Infections and infestations) | 1 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 1 | 2 | 0 | 3
Infected bite (Infections and infestations) | 3 | 2 | 1 | 6
Infected dermal cyst (Infections and infestations) | 1 | 0 | 0 | 1
Infected skin ulcer (Infections and infestations) | 2 | 1 | 0 | 3
Infection (Infections and infestations) | 1 | 1 | 0 | 2
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 18 | 15 | 0 | 33
Injection site cellulitis (Infections and infestations) | 1 | 1 | 0 | 2
Kidney infection (Infections and infestations) | 2 | 2 | 0 | 4
Klebsiella infection (Infections and infestations) | 1 | 0 | 0 | 1
Labyrinthitis (Infections and infestations) | 2 | 1 | 0 | 3
Laryngitis (Infections and infestations) | 5 | 2 | 1 | 8
Localised infection (Infections and infestations) | 3 | 10 | 0 | 13
Lower respiratory tract infection (Infections and infestations) | 29 | 19 | 7 | 55
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 1
Lyme disease (Infections and infestations) | 1 | 2 | 0 | 3
Lymphangitis (Infections and infestations) | 1 | 0 | 0 | 1
Mastitis (Infections and infestations) | 1 | 0 | 0 | 1
Nail bed infection (Infections and infestations) | 0 | 1 | 0 | 1
Nail infection (Infections and infestations) | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 61 | 44 | 5 | 110
Onychomycosis (Infections and infestations) | 12 | 2 | 0 | 14
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 1
Oral fungal infection (Infections and infestations) | 1 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 3 | 0 | 4
Oral infection (Infections and infestations) | 1 | 0 | 0 | 1
Orchitis (Infections and infestations) | 1 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 3 | 0 | 3
Otitis externa (Infections and infestations) | 2 | 6 | 0 | 8
Otitis media (Infections and infestations) | 4 | 3 | 0 | 7
Otitis media acute (Infections and infestations) | 2 | 2 | 0 | 4
Otitis media chronic (Infections and infestations) | 1 | 0 | 0 | 1
Paronychia (Infections and infestations) | 3 | 1 | 0 | 4
Parotitis (Infections and infestations) | 0 | 1 | 0 | 1
Penile infection (Infections and infestations) | 1 | 0 | 0 | 1
Perineal infection (Infections and infestations) | 0 | 1 | 0 | 1
Periodontitis (Infections and infestations) | 3 | 0 | 0 | 3
Pharyngitis (Infections and infestations) | 8 | 2 | 0 | 10
Pharyngitis streptococcal (Infections and infestations) | 2 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 28 | 20 | 2 | 50
Post procedural infection (Infections and infestations) | 0 | 1 | 0 | 1
Post-acute COVID-19 syndrome (Infections and infestations) | 1 | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 1 | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 1
Pulpitis dental (Infections and infestations) | 0 | 2 | 0 | 2
Pyelonephritis (Infections and infestations) | 1 | 1 | 0 | 2
Pyelonephritis chronic (Infections and infestations) | 1 | 0 | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 7 | 9 | 0 | 16
Respiratory tract infection viral (Infections and infestations) | 1 | 1 | 0 | 2
Rhinitis (Infections and infestations) | 7 | 2 | 3 | 12
Root canal infection (Infections and infestations) | 1 | 0 | 0 | 1
Rotavirus infection (Infections and infestations) | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 2 | 1 | 0 | 3
Septic shock (Infections and infestations) | 0 | 1 | 0 | 1
Sinobronchitis (Infections and infestations) | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 14 | 30 | 1 | 45
Sinusitis bacterial (Infections and infestations) | 0 | 2 | 0 | 2
Skin candida (Infections and infestations) | 0 | 1 | 0 | 1
Skin infection (Infections and infestations) | 2 | 2 | 0 | 4
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 5 | 0 | 0 | 5
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 2 | 0 | 0 | 2
Subcutaneous abscess (Infections and infestations) | 4 | 4 | 0 | 8
Suspected COVID-19 (Infections and infestations) | 0 | 4 | 0 | 4
Tick-borne fever (Infections and infestations) | 1 | 0 | 0 | 1
Tinea infection (Infections and infestations) | 0 | 1 | 0 | 1
Tinea pedis (Infections and infestations) | 1 | 1 | 0 | 2
Tonsillitis (Infections and infestations) | 0 | 3 | 1 | 4
Tooth abscess (Infections and infestations) | 8 | 12 | 1 | 21
Tooth infection (Infections and infestations) | 5 | 3 | 1 | 9
Tracheitis (Infections and infestations) | 0 | 2 | 0 | 2
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 56 | 50 | 4 | 110
Urinary tract infection (Infections and infestations) | 77 | 60 | 10 | 147
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 1
Varicella zoster virus infection (Infections and infestations) | 2 | 0 | 0 | 2
Vestibular neuronitis (Infections and infestations) | 0 | 1 | 0 | 1
Viral infection (Infections and infestations) | 8 | 2 | 2 | 12
Viral upper respiratory tract infection (Infections and infestations) | 0 | 3 | 1 | 4
Vulvitis (Infections and infestations) | 1 | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 1 | 1 | 0 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 1 | 2
Wound infection (Infections and infestations) | 1 | 1 | 0 | 2
Accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Administration related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 3 | 2 | 0 | 5
Animal bite (Injury, poisoning and procedural complications) | 2 | 3 | 0 | 5
Animal scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 3 | 4 | 0 | 7
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 5 | 8 | 1 | 14
Arthropod sting (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 3
Avulsion fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Bone contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Burns first degree (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Chest injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 5
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Complications of transplanted lung (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 15 | 21 | 2 | 38
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Costochondral separation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Ear injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Electric shock (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2
Epicondylitis (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 4
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Eye injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 2 | 3 | 0 | 5
Fall (Injury, poisoning and procedural complications) | 33 | 42 | 6 | 81
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Foot fracture (Injury, poisoning and procedural complications) | 3 | 4 | 1 | 8
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Foreign body (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Foreign body in ear (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Foreign body in eye (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Hand fracture (Injury, poisoning and procedural complications) | 8 | 3 | 1 | 12
Head injury (Injury, poisoning and procedural complications) | 4 | 1 | 0 | 5
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 4
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Injection related reaction (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 4
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Intra-ocular injection complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 4 | 7 | 1 | 12
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 8 | 7 | 0 | 15
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 10 | 15 | 1 | 26
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 5 | 2 | 0 | 7
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 3
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 3
Muscle strain (Injury, poisoning and procedural complications) | 7 | 4 | 0 | 11
Musculoskeletal foreign body (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Neck injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Peripancreatic fluid collection (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Post procedural constipation (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Post procedural hypothyroidism (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Post vaccination syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Procedural headache (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 4 | 10 | 3 | 17
Radiation injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Radiation proctitis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 4 | 0 | 4
Rib fracture (Injury, poisoning and procedural complications) | 8 | 8 | 1 | 17
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 5
Skin abrasion (Injury, poisoning and procedural complications) | 7 | 5 | 0 | 12
Skin injury (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 3
Skin laceration (Injury, poisoning and procedural complications) | 18 | 11 | 2 | 31
Skull fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Soft tissue injury (Injury, poisoning and procedural complications) | 6 | 3 | 0 | 9
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 5 | 0 | 8
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 3
Splinter (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 5
Thermal burn (Injury, poisoning and procedural complications) | 4 | 0 | 1 | 5
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 4
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 3
Tobacco poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 2 | 3 | 1 | 6
Traumatic arthrosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 3
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 3
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 5 | 2 | 0 | 7
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 4 | 1 | 0 | 5
Alanine aminotransferase increased (Investigations) | 6 | 4 | 1 | 11
Antiphospholipid antibodies (Investigations) | 0 | 1 | 0 | 1
Aortic bruit (Investigations) | 0 | 1 | 0 | 1
Arteriogram coronary normal (Investigations) | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 5 | 1 | 9
Bilirubin conjugated increased (Investigations) | 0 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 7 | 5 | 0 | 12
Blood bilirubin increased (Investigations) | 6 | 7 | 1 | 14
Blood bilirubin unconjugated increased (Investigations) | 1 | 0 | 0 | 1
Blood calcium decreased (Investigations) | 0 | 1 | 0 | 1
Blood calcium increased (Investigations) | 0 | 0 | 1 | 1
Blood cholesterol increased (Investigations) | 1 | 0 | 0 | 1
Blood creatine abnormal (Investigations) | 1 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 27 | 31 | 0 | 58
Blood creatinine increased (Investigations) | 8 | 7 | 0 | 15
Blood folate decreased (Investigations) | 2 | 4 | 0 | 6
Blood glucose abnormal (Investigations) | 2 | 0 | 0 | 2
Blood glucose increased (Investigations) | 1 | 1 | 3 | 5
Blood homocysteine increased (Investigations) | 1 | 0 | 0 | 1
Blood iron decreased (Investigations) | 1 | 1 | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 1
Blood lactic acid increased (Investigations) | 3 | 0 | 0 | 3
Blood potassium decreased (Investigations) | 1 | 2 | 0 | 3
Blood potassium increased (Investigations) | 2 | 1 | 1 | 4
Blood pressure ambulatory increased (Investigations) | 1 | 0 | 0 | 1
Blood pressure decreased (Investigations) | 1 | 0 | 0 | 1
Blood pressure diastolic decreased (Investigations) | 0 | 1 | 0 | 1
Blood pressure increased (Investigations) | 13 | 14 | 0 | 27
Blood pressure systolic increased (Investigations) | 2 | 0 | 0 | 2
Blood sodium decreased (Investigations) | 1 | 2 | 0 | 3
Blood sodium increased (Investigations) | 1 | 0 | 0 | 1
Blood testosterone decreased (Investigations) | 1 | 1 | 0 | 2
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 0 | 1
Blood triglycerides increased (Investigations) | 4 | 8 | 1 | 13
Blood urea increased (Investigations) | 1 | 1 | 0 | 2
Blood urine present (Investigations) | 2 | 2 | 0 | 4
Body temperature abnormal (Investigations) | 1 | 0 | 0 | 1
Borrelia test positive (Investigations) | 0 | 1 | 0 | 1
Brain natriuretic peptide increased (Investigations) | 3 | 2 | 0 | 5
C-reactive protein increased (Investigations) | 8 | 7 | 2 | 17
Carbohydrate antigen 15-3 increased (Investigations) | 0 | 1 | 0 | 1
Cardiac murmur (Investigations) | 5 | 5 | 0 | 10
Cardiac stress test abnormal (Investigations) | 3 | 0 | 0 | 3
Carotid bruit (Investigations) | 0 | 1 | 0 | 1
Coronavirus test positive (Investigations) | 1 | 4 | 3 | 8
Ejection fraction decreased (Investigations) | 0 | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 1 | 0 | 2
Electrocardiogram ST-T change (Investigations) | 1 | 0 | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 2 | 0 | 0 | 2
Electrocardiogram abnormal (Investigations) | 4 | 1 | 0 | 5
Electrocardiogram repolarisation abnormality (Investigations) | 0 | 1 | 0 | 1
Fibrin D dimer increased (Investigations) | 1 | 1 | 0 | 2
Gamma-glutamyltransferase abnormal (Investigations) | 1 | 1 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 16 | 23 | 0 | 39
Glomerular filtration rate decreased (Investigations) | 9 | 8 | 1 | 18
Glucose urine present (Investigations) | 1 | 0 | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 13 | 15 | 1 | 29
Haematology test abnormal (Investigations) | 0 | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 3 | 2 | 1 | 6
Haemoglobin increased (Investigations) | 1 | 0 | 0 | 1
Heart rate decreased (Investigations) | 1 | 0 | 0 | 1
Heart rate irregular (Investigations) | 2 | 3 | 0 | 5
Helicobacter test positive (Investigations) | 0 | 1 | 0 | 1
Hepatic enzyme abnormal (Investigations) | 0 | 1 | 0 | 1
Hepatic enzyme increased (Investigations) | 9 | 7 | 1 | 17
Immunoglobulins decreased (Investigations) | 1 | 0 | 0 | 1
Immunoglobulins increased (Investigations) | 0 | 1 | 0 | 1
International normalised ratio increased (Investigations) | 2 | 2 | 0 | 4
Intraocular pressure increased (Investigations) | 2 | 0 | 0 | 2
Laboratory test abnormal (Investigations) | 0 | 1 | 0 | 1
Lipase increased (Investigations) | 2 | 0 | 0 | 2
Lipids increased (Investigations) | 0 | 1 | 0 | 1
Lipoprotein (a) increased (Investigations) | 0 | 0 | 1 | 1
Lipoprotein increased (Investigations) | 0 | 0 | 1 | 1
Liver function test abnormal (Investigations) | 0 | 6 | 1 | 7
Liver function test increased (Investigations) | 2 | 7 | 0 | 9
Low density lipoprotein increased (Investigations) | 5 | 3 | 0 | 8
Mean cell volume increased (Investigations) | 1 | 1 | 0 | 2
Monofilament pressure perception test abnormal (Investigations) | 1 | 0 | 0 | 1
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 1 | 0 | 1
Nitrite urine (Investigations) | 0 | 1 | 0 | 1
Occult blood positive (Investigations) | 2 | 0 | 0 | 2
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0 | 1
Prostatic specific antigen increased (Investigations) | 3 | 1 | 0 | 4
Protein urine present (Investigations) | 0 | 1 | 0 | 1
Respiratory rate increased (Investigations) | 0 | 1 | 0 | 1
Romberg test positive (Investigations) | 1 | 0 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 1 | 2 | 1 | 4
Scan myocardial perfusion abnormal (Investigations) | 2 | 0 | 0 | 2
Serum ferritin decreased (Investigations) | 2 | 0 | 0 | 2
Serum ferritin increased (Investigations) | 0 | 1 | 0 | 1
Thyroxine increased (Investigations) | 0 | 1 | 0 | 1
Transaminases increased (Investigations) | 0 | 2 | 0 | 2
Troponin increased (Investigations) | 3 | 5 | 0 | 8
Tryptase increased (Investigations) | 1 | 0 | 0 | 1
Ultrasound Doppler abnormal (Investigations) | 0 | 0 | 1 | 1
Ultrasound scan abnormal (Investigations) | 1 | 0 | 0 | 1
Urinary system x-ray abnormal (Investigations) | 0 | 1 | 0 | 1
Urine analysis abnormal (Investigations) | 3 | 1 | 0 | 4
Urine output decreased (Investigations) | 0 | 1 | 0 | 1
Vitamin D decreased (Investigations) | 1 | 1 | 0 | 2
Weight decreased (Investigations) | 12 | 7 | 0 | 19
Weight increased (Investigations) | 4 | 2 | 0 | 6
White blood cell count increased (Investigations) | 0 | 1 | 0 | 1
White blood cells urine positive (Investigations) | 1 | 0 | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Carbohydrate intolerance (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 4 | 4 | 0 | 8
Dehydration (Metabolism and nutrition disorders) | 10 | 11 | 0 | 21
Diabetes mellitus (Metabolism and nutrition disorders) | 98 | 100 | 7 | 205
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 114 | 109 | 3 | 226
Diabetic complication (Metabolism and nutrition disorders) | 0 | 3 | 0 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 4 | 4 | 0 | 8
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 1 | 0 | 3
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Folate deficiency (Metabolism and nutrition disorders) | 2 | 3 | 0 | 5
Fructose intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 15 | 10 | 0 | 25
Gout (Metabolism and nutrition disorders) | 15 | 21 | 1 | 37
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 9 | 1 | 16
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 8 | 1 | 17
Hyperlipidaemia (Metabolism and nutrition disorders) | 7 | 4 | 1 | 12
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 10 | 6 | 0 | 16
Hyperuricaemia (Metabolism and nutrition disorders) | 9 | 7 | 0 | 16
Hypervitaminosis D (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 3 | 0 | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 4 | 1 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 19 | 13 | 0 | 32
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 2 | 0 | 10
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 5 | 1 | 11
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 4
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Impaired fasting glucose (Metabolism and nutrition disorders) | 4 | 2 | 0 | 6
Insulin resistance (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Iron deficiency (Metabolism and nutrition disorders) | 5 | 2 | 0 | 7
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
Latent autoimmune diabetes in adults (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Magnesium deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 5 | 0 | 6
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 2 | 1 | 0 | 3
Overweight (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Postprandial hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 32 | 41 | 4 | 77
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 6 | 3 | 0 | 9
Vitamin D deficiency (Metabolism and nutrition disorders) | 14 | 15 | 1 | 30
Ankle impingement (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 94 | 102 | 5 | 201
Arthritis (Musculoskeletal and connective tissue disorders) | 14 | 12 | 2 | 28
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 67 | 51 | 8 | 126
Bone atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 4 | 6 | 3 | 13
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 3
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Chronic kidney disease-mineral and bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 4
Degenerative bone disease (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Diffuse idiopathic skeletal hyperostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 3 | 5 | 0 | 8
Exostosis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 5
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0 | 7
Foot deformity (Musculoskeletal and connective tissue disorders) | 4 | 4 | 1 | 9
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0 | 7
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 6 | 5 | 0 | 11
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 5 | 4 | 1 | 10
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 7 | 9 | 1 | 17
Joint effusion (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | 6
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 6 | 5 | 1 | 12
Ligament calcification (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 4
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1 | 8
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 4
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscle oedema (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 26 | 10 | 1 | 37
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 8 | 4 | 1 | 13
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1 | 8
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 19 | 26 | 3 | 48
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 16 | 14 | 1 | 31
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 60 | 53 | 6 | 119
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 6
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 | 8 | 2 | 13
Osteoporosis postmenopausal (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 43 | 38 | 5 | 86
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 4
Periostitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 9 | 4 | 1 | 14
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 5 | 4 | 0 | 9
Rib deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 14 | 14 | 2 | 30
SLE arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Sacroiliac joint dysfunction (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 12 | 15 | 2 | 29
Spinal pain (Musculoskeletal and connective tissue disorders) | 4 | 7 | 0 | 11
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 3
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 7 | 5 | 0 | 12
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 3
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 4
Tendonitis (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2 | 9
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 4
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 10 | 7 | 1 | 18
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1 | 4
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24 | 5 | 1 | 30
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Benign laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 4
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Eye naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 4
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 3
Juvenile melanoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0 | 4
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2 | 0 | 7
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Oesophageal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 2
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 0 | 7
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Renal hamartoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4 | 3 | 12
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 3
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 4
Skin squamous cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1 | 4
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Vulvovaginal warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Ageusia (Nervous system disorders) | 0 | 2 | 0 | 2
Akinesia (Nervous system disorders) | 0 | 1 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 1 | 1
Amnesia (Nervous system disorders) | 6 | 3 | 0 | 9
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 1
Arachnoid cyst (Nervous system disorders) | 1 | 1 | 0 | 2
Balance disorder (Nervous system disorders) | 8 | 2 | 1 | 11
Bell's palsy (Nervous system disorders) | 2 | 1 | 1 | 4
Burning sensation (Nervous system disorders) | 1 | 2 | 0 | 3
Carotid arteriosclerosis (Nervous system disorders) | 3 | 2 | 1 | 6
Carotid artery disease (Nervous system disorders) | 2 | 0 | 0 | 2
Carotid artery occlusion (Nervous system disorders) | 0 | 1 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 6 | 4 | 0 | 10
Carpal tunnel syndrome (Nervous system disorders) | 13 | 8 | 1 | 22
Cerebellar atrophy (Nervous system disorders) | 0 | 1 | 0 | 1
Cerebral arteriosclerosis (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebral atrophy (Nervous system disorders) | 2 | 1 | 1 | 4
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 1
Cerebral microangiopathy (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebral small vessel ischaemic disease (Nervous system disorders) | 0 | 2 | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 3 | 0 | 0 | 3
Cervical radiculopathy (Nervous system disorders) | 6 | 2 | 0 | 8
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0 | 1
Cervicogenic headache (Nervous system disorders) | 1 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 4 | 2 | 0 | 6
Cortical laminar necrosis (Nervous system disorders) | 0 | 1 | 0 | 1
Cubital tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 1
Dementia (Nervous system disorders) | 3 | 2 | 0 | 5
Dementia Alzheimer's type (Nervous system disorders) | 2 | 2 | 0 | 4
Diabetic neuropathy (Nervous system disorders) | 6 | 4 | 1 | 11
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 40 | 42 | 6 | 88
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 1
Encephalopathy (Nervous system disorders) | 3 | 0 | 0 | 3
Epilepsy (Nervous system disorders) | 2 | 1 | 0 | 3
Essential tremor (Nervous system disorders) | 0 | 2 | 0 | 2
Facial paralysis (Nervous system disorders) | 0 | 2 | 0 | 2
Facial paresis (Nervous system disorders) | 1 | 0 | 0 | 1
Head discomfort (Nervous system disorders) | 1 | 0 | 1 | 2
Headache (Nervous system disorders) | 41 | 37 | 5 | 83
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 5 | 7 | 0 | 12
Hyporeflexia (Nervous system disorders) | 1 | 2 | 0 | 3
Hyposmia (Nervous system disorders) | 0 | 1 | 0 | 1
Intercostal neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0 | 1
Intracranial mass (Nervous system disorders) | 1 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 1
Lethargy (Nervous system disorders) | 2 | 1 | 0 | 3
Loss of consciousness (Nervous system disorders) | 1 | 1 | 0 | 2
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 1 | 2
Lumbosacral radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 5 | 2 | 1 | 8
Migraine (Nervous system disorders) | 5 | 1 | 0 | 6
Morton's neuralgia (Nervous system disorders) | 2 | 0 | 0 | 2
Muscle contractions involuntary (Nervous system disorders) | 0 | 1 | 0 | 1
Myelopathy (Nervous system disorders) | 0 | 0 | 1 | 1
Nerve compression (Nervous system disorders) | 3 | 5 | 0 | 8
Neuralgia (Nervous system disorders) | 3 | 3 | 0 | 6
Neuropathy peripheral (Nervous system disorders) | 18 | 11 | 4 | 33
Pachymeningitis (Nervous system disorders) | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 6 | 4 | 2 | 12
Paralysis (Nervous system disorders) | 0 | 2 | 0 | 2
Parkinson's disease (Nervous system disorders) | 5 | 3 | 0 | 8
Partial seizures (Nervous system disorders) | 1 | 0 | 0 | 1
Periodic limb movement disorder (Nervous system disorders) | 1 | 0 | 0 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 1 | 1 | 0 | 2
Polyneuropathy (Nervous system disorders) | 2 | 1 | 0 | 3
Post herpetic neuralgia (Nervous system disorders) | 1 | 1 | 0 | 2
Post polio syndrome (Nervous system disorders) | 1 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 6 | 4 | 1 | 11
Quadrantanopia (Nervous system disorders) | 0 | 0 | 1 | 1
Radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 1 | 1 | 0 | 2
Sciatica (Nervous system disorders) | 15 | 22 | 1 | 38
Seizure (Nervous system disorders) | 4 | 2 | 0 | 6
Senile dementia (Nervous system disorders) | 0 | 1 | 0 | 1
Sensory disturbance (Nervous system disorders) | 0 | 1 | 0 | 1
Sensory loss (Nervous system disorders) | 1 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 1 | 0 | 1
Spinal claudication (Nervous system disorders) | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 16 | 15 | 0 | 31
Taste disorder (Nervous system disorders) | 3 | 0 | 0 | 3
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 1
Thoracic radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 1
Thunderclap headache (Nervous system disorders) | 1 | 0 | 0 | 1
Transient global amnesia (Nervous system disorders) | 1 | 0 | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 2 | 2 | 0 | 4
Tremor (Nervous system disorders) | 7 | 4 | 1 | 12
Trigeminal neuralgia (Nervous system disorders) | 2 | 1 | 0 | 3
Ulnar neuritis (Nervous system disorders) | 0 | 0 | 1 | 1
VIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0 | 1
Vascular dementia (Nervous system disorders) | 2 | 1 | 0 | 3
Vascular encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 1
Vascular parkinsonism (Nervous system disorders) | 1 | 0 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0 | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 0 | 1 | 0 | 1
Device dislocation (Product Issues) | 0 | 2 | 0 | 2
Device malfunction (Product Issues) | 0 | 1 | 0 | 1
Device physical property issue (Product Issues) | 1 | 0 | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0 | 1
Acute stress disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 3 | 0 | 3
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 2 | 0 | 2
Alcoholism (Psychiatric disorders) | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 16 | 21 | 1 | 38
Anxiety disorder (Psychiatric disorders) | 2 | 0 | 0 | 2
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 | 1 | 0 | 2
Bipolar II disorder (Psychiatric disorders) | 1 | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 6 | 1 | 0 | 7
Delirium (Psychiatric disorders) | 2 | 2 | 0 | 4
Delusion (Psychiatric disorders) | 0 | 2 | 0 | 2
Depressed mood (Psychiatric disorders) | 5 | 4 | 0 | 9
Depression (Psychiatric disorders) | 29 | 19 | 3 | 51
Grief reaction (Psychiatric disorders) | 1 | 1 | 0 | 2
Habit cough (Psychiatric disorders) | 0 | 1 | 0 | 1
Hallucination (Psychiatric disorders) | 4 | 0 | 0 | 4
Hallucination, visual (Psychiatric disorders) | 0 | 3 | 0 | 3
Initial insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 13 | 15 | 0 | 28
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 1
Libido decreased (Psychiatric disorders) | 0 | 1 | 0 | 1
Loss of libido (Psychiatric disorders) | 1 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 1 | 0 | 3
Nightmare (Psychiatric disorders) | 0 | 1 | 0 | 1
Obsessive-compulsive disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1 | 1 | 2
Poor quality sleep (Psychiatric disorders) | 0 | 1 | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 1 | 1
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 1
Schizoaffective disorder bipolar type (Psychiatric disorders) | 1 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 3 | 5 | 0 | 8
Stress (Psychiatric disorders) | 1 | 3 | 0 | 4
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 11 | 18 | 0 | 29
Albuminuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0 | 0 | 1
Bladder disorder (Renal and urinary disorders) | 1 | 0 | 0 | 1
Bladder diverticulum (Renal and urinary disorders) | 0 | 1 | 0 | 1
Bladder irritation (Renal and urinary disorders) | 1 | 0 | 0 | 1
Bladder outlet obstruction (Renal and urinary disorders) | 1 | 2 | 0 | 3
Bladder prolapse (Renal and urinary disorders) | 1 | 0 | 0 | 1
Bladder stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 23 | 20 | 1 | 44
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0 | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 1 | 2 | 0 | 3
Diabetic nephropathy (Renal and urinary disorders) | 1 | 2 | 0 | 3
Dysuria (Renal and urinary disorders) | 6 | 2 | 2 | 10
End stage renal disease (Renal and urinary disorders) | 2 | 1 | 0 | 3
Genitourinary symptom (Renal and urinary disorders) | 0 | 1 | 0 | 1
Glycosuria (Renal and urinary disorders) | 2 | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 14 | 13 | 0 | 27
Hydronephrosis (Renal and urinary disorders) | 2 | 0 | 0 | 2
Hypertensive nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 5 | 6 | 0 | 11
Leukocyturia (Renal and urinary disorders) | 1 | 2 | 0 | 3
Lower urinary tract symptoms (Renal and urinary disorders) | 1 | 3 | 0 | 4
Microalbuminuria (Renal and urinary disorders) | 3 | 1 | 0 | 4
Micturition urgency (Renal and urinary disorders) | 1 | 1 | 1 | 3
Nephritic syndrome (Renal and urinary disorders) | 0 | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 15 | 10 | 1 | 26
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 1
Neurogenic bladder (Renal and urinary disorders) | 0 | 1 | 0 | 1
Nocturia (Renal and urinary disorders) | 3 | 1 | 0 | 4
Pollakiuria (Renal and urinary disorders) | 6 | 4 | 0 | 10
Polyuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 4 | 2 | 0 | 6
Pyelocaliectasis (Renal and urinary disorders) | 0 | 1 | 0 | 1
Renal aneurysm (Renal and urinary disorders) | 0 | 1 | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 1 | 1 | 2
Renal colic (Renal and urinary disorders) | 4 | 2 | 0 | 6
Renal cyst (Renal and urinary disorders) | 9 | 22 | 0 | 31
Renal disorder (Renal and urinary disorders) | 1 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 5 | 6 | 0 | 11
Renal impairment (Renal and urinary disorders) | 24 | 30 | 0 | 54
Renal mass (Renal and urinary disorders) | 1 | 0 | 0 | 1
Renal necrosis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Renal pain (Renal and urinary disorders) | 1 | 0 | 0 | 1
Strangury (Renal and urinary disorders) | 0 | 1 | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 4 | 0 | 0 | 4
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 2 | 0 | 2
Urethral stenosis (Renal and urinary disorders) | 0 | 2 | 0 | 2
Urge incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 6 | 5 | 1 | 12
Urinary retention (Renal and urinary disorders) | 5 | 4 | 0 | 9
Urinary tract disorder (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary tract inflammation (Renal and urinary disorders) | 2 | 0 | 0 | 2
Urine odour abnormal (Renal and urinary disorders) | 0 | 1 | 0 | 1
Acquired phimosis (Reproductive system and breast disorders) | 2 | 0 | 0 | 2
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 | 2 | 0 | 3
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 26 | 20 | 2 | 48
Breast disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 2 | 0 | 2
Breast necrosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 11 | 8 | 2 | 21
Genital prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 3 | 1 | 4
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Nipple exudate bloody (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Ovarian calcification (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Ovarian mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 1 | 0 | 2
Penile discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Peyronie's disease (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Prostatic mass (Reproductive system and breast disorders) | 0 | 1 | 1 | 2
Prostatism (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 2 | 6 | 1 | 9
Prostatomegaly (Reproductive system and breast disorders) | 6 | 5 | 0 | 11
Rectocele (Reproductive system and breast disorders) | 1 | 1 | 0 | 2
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Sexual dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Spermatocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Testicular hypertrophy (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Testicular mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 2 | 1 | 0 | 3
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Vulva cyst (Reproductive system and breast disorders) | 2 | 0 | 1 | 3
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Vulvovaginal inflammation (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 1 | 0 | 2
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 6
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 10 | 5 | 2 | 17
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 5
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 4
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 13 | 24 | 2 | 39
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 32 | 3 | 71
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 39 | 31 | 6 | 76
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 11 | 9 | 3 | 23
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Epiglottic oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 6 | 0 | 16
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 4
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Laryngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 3
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 4
Nasal mucosal blistering (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 1 | 13
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 12 | 1 | 18
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 3
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 0 | 7
Pulmonary calcification (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0 | 6
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 3
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 0 | 13
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 4
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 0 | 11
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 5
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 6
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 0 | 8
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 1 | 8
Vocal cord cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 5 | 4 | 2 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 5
Alopecia areata (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 3
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Blister (Skin and subcutaneous tissue disorders) | 4 | 3 | 0 | 7
Cutaneous calcification (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 4
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 3 | 1 | 6
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 | 3 | 0 | 6
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 3
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 4
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 5
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 6 | 7 | 1 | 14
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2 | 5 | 10
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 3 | 0 | 8
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 3
Hypertrophic scar (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 3
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Lentigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Milia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Pemphigus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pityriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Polymorphic light eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 7 | 1 | 16
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 6 | 2 | 0 | 8
Purpura senile (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 13 | 9 | 1 | 23
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 3
Reactive perforating collagenosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 5
Sebaceous hyperplasia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Sensitive skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Skin fibrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Skin indentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 6 | 7 | 1 | 14
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Skin texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 6 | 6 | 1 | 13
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 4
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 5
Xanthoma (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Family stress (Social circumstances) | 0 | 1 | 0 | 1
Aneurysm (Vascular disorders) | 1 | 0 | 0 | 1
Angiodysplasia (Vascular disorders) | 0 | 1 | 0 | 1
Angiopathy (Vascular disorders) | 0 | 1 | 0 | 1
Aortic aneurysm (Vascular disorders) | 2 | 4 | 0 | 6
Aortic aneurysm rupture (Vascular disorders) | 0 | 1 | 0 | 1
Aortic arteriosclerosis (Vascular disorders) | 2 | 2 | 0 | 4
Aortic dilatation (Vascular disorders) | 2 | 3 | 0 | 5
Aortic stenosis (Vascular disorders) | 6 | 3 | 1 | 10
Arterial occlusive disease (Vascular disorders) | 1 | 1 | 0 | 2
Arterial thrombosis (Vascular disorders) | 0 | 1 | 0 | 1
Arteriosclerosis (Vascular disorders) | 8 | 2 | 0 | 10
Arteritis (Vascular disorders) | 1 | 0 | 0 | 1
Blood pressure fluctuation (Vascular disorders) | 1 | 0 | 0 | 1
Blood pressure inadequately controlled (Vascular disorders) | 2 | 2 | 0 | 4
Circulatory collapse (Vascular disorders) | 0 | 2 | 0 | 2
Cyanosis (Vascular disorders) | 0 | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 5 | 2 | 0 | 7
Diastolic hypertension (Vascular disorders) | 1 | 0 | 0 | 1
Essential hypertension (Vascular disorders) | 0 | 1 | 0 | 1
Extravasation blood (Vascular disorders) | 0 | 1 | 0 | 1
Flushing (Vascular disorders) | 0 | 1 | 0 | 1
Haematoma (Vascular disorders) | 3 | 3 | 1 | 7
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 4 | 0 | 4
Hypertension (Vascular disorders) | 106 | 110 | 9 | 225
Hypertensive crisis (Vascular disorders) | 3 | 2 | 0 | 5
Hypertensive urgency (Vascular disorders) | 0 | 2 | 0 | 2
Hypotension (Vascular disorders) | 21 | 21 | 1 | 43
Iliac artery arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 1
Iliac artery stenosis (Vascular disorders) | 1 | 1 | 0 | 2
Intermittent claudication (Vascular disorders) | 0 | 5 | 3 | 8
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 3 | 0 | 1 | 4
Microangiopathy (Vascular disorders) | 0 | 1 | 0 | 1
Orthostatic hypertension (Vascular disorders) | 1 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 3 | 5 | 0 | 8
Peripheral arterial occlusive disease (Vascular disorders) | 11 | 10 | 1 | 22
Peripheral artery occlusion (Vascular disorders) | 2 | 5 | 0 | 7
Peripheral artery stenosis (Vascular disorders) | 1 | 1 | 0 | 2
Peripheral coldness (Vascular disorders) | 0 | 1 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 2 | 0 | 2
Peripheral vascular disorder (Vascular disorders) | 5 | 2 | 0 | 7
Peripheral venous disease (Vascular disorders) | 6 | 8 | 0 | 14
Phlebitis (Vascular disorders) | 1 | 1 | 0 | 2
Phlebitis deep (Vascular disorders) | 0 | 1 | 0 | 1
Phlebitis superficial (Vascular disorders) | 0 | 1 | 0 | 1
Post thrombotic syndrome (Vascular disorders) | 1 | 1 | 0 | 2
Raynaud's phenomenon (Vascular disorders) | 1 | 2 | 0 | 3
Superficial vein prominence (Vascular disorders) | 0 | 1 | 0 | 1
Superficial vein thrombosis (Vascular disorders) | 0 | 2 | 0 | 2
Systolic hypertension (Vascular disorders) | 0 | 1 | 0 | 1
Thrombophlebitis (Vascular disorders) | 3 | 2 | 0 | 5
Thrombosed varicose vein (Vascular disorders) | 1 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 1
Varicose vein (Vascular disorders) | 6 | 9 | 0 | 15
Vasculitis (Vascular disorders) | 0 | 1 | 0 | 1
Venous hypertension (Vascular disorders) | 0 | 1 | 0 | 1
White coat hypertension (Vascular disorders) | 0 | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT03814187/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-04): https://cdn.clinicaltrials.gov/large-docs/87/NCT03814187/SAP_001.pdf